CLINICAL TRIAL: NCT01327846
Title: A Randomized, Double-blind, Placebo-controlled, Event-driven Trial of Quarterly Subcutaneous Canakinumab in the Prevention of Recurrent Cardiovascular Events Among Stable Post-myocardial Infarction Patients With Elevated hsCRP
Brief Title: Cardiovascular Risk Reduction Study (Reduction in Recurrent Major CV Disease Events)
Acronym: CANTOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CACZ885M2301; 2010-022970-14 (EudraCT Number)
Record Dates: First submitted 2011-03-29; First posted 2011-04-04 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Atherosclerosis
Keywords: Cardiovascular Death; Myocardial Infarction; Stroke; Canakinumab; IL-1B; hsCRP
MeSH Terms: conditions — Atherosclerosis; Myocardial Infarction; Stroke | interventions — canakinumab; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Canakinumab Dose 50 mg (Experimental): Pivotal Phase:
  Blinded Canakinumab 50 mg quarterly subcutaneous + standard of care therapy.
  Extension Phase:
  Switched to open-label Canakinumab 150 mg quarterly subcutaneous + standard of care therapy
  Interventions: Drug: Canakinumab; Drug: Standard of care
- Canakinumab Dose 150 mg (Experimental): Pivotal Phase:
  Switched to open-label Canakinumab 150 mg quarterly subcutaneous + standard of care therapy
  Interventions: Drug: Canakinumab; Drug: Standard of care
- Canakinumab Dose 300 mg (Experimental): Pivotal Phase:
  Blinded Canakinumab 300 mg quarterly subcutaneous (with one additional dose at week 2) + standard of care therapy.
  Extension phase:
  Switched to open-label Canakinumab 150 mg quarterly subcutaneous + standard of care therapy
  Interventions: Drug: Canakinumab; Drug: Standard of care
- Placebo (Placebo Comparator): Pivotal Phase:
  Blinded matching placebo quarterly subcutaneous + standard of care therapy.
  Extension Phase:
  Switched to open-label Canakinumab 150 mg quarterly subcutaneous + standard of care therapy
  Interventions: Drug: Placebo; Drug: Standard of care

INTERVENTIONS:
Drug: Canakinumab
  Other Names: ACZ885
  Arms: Canakinumab Dose 150 mg; Canakinumab Dose 300 mg; Canakinumab Dose 50 mg
Drug: Placebo
  Arms: Placebo
Drug: Standard of care — Standard of care post-MI background therapy includes, but is not limited to, lipid lowering, anti-hypertensive, beta blockers, and anti-platelet therapy as appropriate

SUMMARY:
Main Study (CACZ885M2301): The purpose of the pivotal phase of this trial was to test the hypothesis that canakinumab treatment of patients with myocardial infarction (MI) at least one month prior to study entry and elevated hsCRP could prevent recurrent cardiovascular events.

The purpose of the extension phase of the main study is to collect additional long-term safety data on continued exposure to canakinumab in patients who participated in the pivotal phase.

Sub-study 1 (CACZ885M2301S1): The purpose of this sub-study was to evaluate the effect of quarterly subcutaneous canakinumab treatment for 24 months comparted with placebo on the carotid plaque burden measured by integrated vascular MRI in patients enrolled in the CACZ885M2301 study (CANTOS).

Sub-study 2 (CACZ885M2301S2): The purpose of this CANTOS sub-study was to determine whether, in patients with type 2 diabetes participating in the CANTOS main study, canakinumab compared to placebo, on top of standard of care could increase insulin secretion and insulin sensitivity.

DETAILED DESCRIPTION:
Sub-study 1 and 2 were terminated prior to data collection from subjects. However, there is an ongoing extension trial where patients are receiving open-drug label.

ELIGIBILITY:
Main Study Inclusion Criteria:

* Written informed consent
* Male, or Female of non-child-bearing potential
* Age ≥ 18 years.
* Spontaneous MI at least 30 days before randomization. hsCRP ≥ 2 mg/L

Substudy 1 Inclusion:

* All Inclusion from Main Study
* Acquisition of evaluable baseline MRI images of bilateral carotid arteries by the imaging core laboratory

Substudy 2 Inclusion:

* All inclusion from Main Study
* T2D at baseline per Main protocol criteria and be on a stable anti-hyperglycemic medication for at least 4 weeks prior to the baseline OGTT test
* Willing to have the OGTT assessment started before 10 am

Main Study Exclusion Criteria:

* Pregnant or nursing (lactating) women
* Women of child-bearing potential
* Any of the following concomitant diseases
* Planned coronary revascularization (PCI or CABG)
* Major non-cardiac surgical or endoscopic procedure within past 6 months
* Multi-vessel CABG surgery within the past 3 years
* Symptomatic patients with Class IV heart failure (HF) (New York Heart Association [NYHA].
* Uncontrolled hypertension
* Uncontrolled diabetes
* History or evidence of active tuberculosis (TB) infection Substudy 1 Exclusion
* All Main exclusion
* Patients with prior history of carotid angioplasty, stenting, or carotid atherectomy
* Patients with contraindications to MRI examination (brain aneurysm clip, implanted neural stimulator, implanted cardiac pacemaker, pacemaker wires or defibrillator, prosthetic heart valves, cochlear implant, ocular foreign body or other implanted body, tattoos, implanted insulin pump, metal shrapnel or bullet)
* Patients prone to claustrophobia or known anxiety disorders
* BMI > 40 kg/m2 Substudy 2 Exclusion
* This sub-study does not have any additional exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10066 (Actual)
Dates: Start 2011-04-11 (Actual); Primary Completion 2017-03-28 (Actual); Study Completion 2019-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (869):
- United States (251):
  - Novartis Investigative Site, Athens, Alabama
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Fairhope, Alabama
  - Novartis Investigative Site, Huntsville, Alabama
  - Novartis Investigative Site, Mobile, Alabama
  - Novartis Investigative Site, Anchorage, Alaska
  - Novartis Investigative Site, Chandler, Arizona
  - Novartis Investigative Site, Glendale, Arizona
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Hot Springs, Arkansas
  - Novartis Investigative Site, Jonesboro, Arkansas
  - Novartis Investigative Site, Little Rock, Arkansas
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Carmichael, California
  - Novartis Investigative Site, Escondido, California
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, Lancaster, California
  - Novartis Investigative Site, Loma Linda, California
  - Novartis Investigative Site, Long Beach, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Los Gatos, California
  - Novartis Investigative Site, Mission Viejo, California
  - Novartis Investigative Site, Newport Beach, California
  - Novartis Investigative Site, Northridge, California
  - Novartis Investigative Site, Oceanside, California
  - Novartis Investigative Site, Orangevale, California
  - Novartis Investigative Site, Palm Springs, California
  - Novartis Investigative Site, Pasadena, California
  - Novartis Investigative Site, Pomona, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Santa Ana, California
  - Novartis Investigative Site, Santa Rosa, California
  - Novartis Investigative Site, Torrance, California
  - Novartis Investigative Site, Tustin, California
  - Novartis Investigative Site, Visalia, California
  - Novartis Investigative Site, Walnut Creek, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Colorado Springs, Colorado
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Norwich, Connecticut
  - Novartis Investigative Site, Newark, Delaware
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Clearwater, Florida
  - Novartis Investigative Site, Coral Springs, Florida
  - Novartis Investigative Site, Davie, Florida
  - Novartis Investigative Site, Daytona Beach, Florida
  - Novartis Investigative Site, DeFuniak Springs, Florida
  - Novartis Investigative Site, Doral, Florida
  - Novartis Investigative Site, Hialeah, Florida
  - Novartis Investigative Site, Hollywood, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Jacksonville Beach, Florida
  - Novartis Investigative Site, Jupiter, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Miami Beach, Florida
  - Novartis Investigative Site, Naples, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Pembroke Pines, Florida
  - Novartis Investigative Site, Pinellas Park, Florida
  - Novartis Investigative Site, Port Charlotte, Florida
  - Novartis Investigative Site, Port Orange, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, South Miami, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Wellington, Florida
  - Novartis Investigative Site, Athens, Georgia
  - Novartis Investigative Site, Augusta, Georgia
  - Novartis Investigative Site, Covington, Georgia
  - Novartis Investigative Site, Cumming, Georgia
  - Novartis Investigative Site, Decatur, Georgia
  - Novartis Investigative Site, Duluth, Georgia
  - Novartis Investigative Site, Macon, Georgia
  - Novartis Investigative Site, Roswell, Georgia
  - Novartis Investigative Site, Savannah, Georgia
  - Novartis Investigative Site, Thomasville, Georgia
  - Novartis Investigative Site, Honolulu, Hawaii
  - Novartis Investigative Site, Coeur d'Alene, Idaho
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Jerseyville, Illinois
  - Novartis Investigative Site, Lombard, Illinois
  - Novartis Investigative Site, Melrose Park, Illinois
  - Novartis Investigative Site, Peoria, Illinois
  - Novartis Investigative Site, Evansville, Indiana
  - Novartis Investigative Site, Ames, Iowa
  - Novartis Investigative Site, Waterloo, Iowa
  - Novartis Investigative Site, Kansas City, Kansas
  - Novartis Investigative Site, Overland Park, Kansas
  - Novartis Investigative Site, Topeka, Kansas
  - Novartis Investigative Site, Wichita, Kansas
  - Novartis Investigative Site, Lexington, Kentucky
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, Madisonville, Kentucky
  - Novartis Investigative Site, Owensboro, Kentucky
  - Novartis Investigative Site, Baton Rouge, Louisiana
  - Novartis Investigative Site, Covington, Louisiana
  - Novartis Investigative Site, Houma, Louisiana
  - Novartis Investigative Site, Lafayette, Louisiana
  - Novartis Investigative Site, Mandeville, Louisiana
  - Novartis Investigative Site, Metairie, Louisiana
  - Novartis Investigative Site, Minden, Louisiana
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Opelousas, Louisiana
  - Novartis Investigative Site, Shreveport, Louisiana
  - Novartis Investigative Site, Slidell, Louisiana
  - Novartis Investigative Site, Winnsboro, Louisiana
  - Novartis Investigative Site, Zachary, Louisiana
  - Novartis Investigative Site, Portland, Maine
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Beltsville, Maryland
  - Novartis Investigative Site, Columbia, Maryland
  - Novartis Investigative Site, Burlington, Massachusetts
  - Novartis Investigative Site, Fall River, Massachusetts
  - Novartis Investigative Site, Haverhill, Massachusetts
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Chelsea, Michigan
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Grand Blanc, Michigan
  - Novartis Investigative Site, Kalamazoo, Michigan
  - Novartis Investigative Site, Midland, Michigan
  - Novartis Investigative Site, Novi, Michigan
  - Novartis Investigative Site, Petoskey, Michigan
  - Novartis Investigative Site, Royal Oak, Michigan
  - Novartis Investigative Site, Saginaw, Michigan
  - Novartis Investigative Site, Wyoming, Michigan
  - Novartis Investigative Site, Bloomington, Minnesota
  - Novartis Investigative Site, Duluth, Minnesota
  - Novartis Investigative Site, Edina, Minnesota
  - Novartis Investigative Site, Fridley, Minnesota
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Robbinsdale, Minnesota
  - Novartis Investigative Site, Saint Cloud, Minnesota
  - Novartis Investigative Site, Saint Paul, Minnesota
  - Novartis Investigative Site, Hattiesburg, Mississippi
  - Novartis Investigative Site, Jackson, Mississippi
  - Novartis Investigative Site, Picayune, Mississippi
  - Novartis Investigative Site, Columbia, Missouri
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, Springfield, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Grand Island, Nebraska
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Nashua, New Hampshire
  - Novartis Investigative Site, Camden, New Jersey
  - Novartis Investigative Site, Freehold, New Jersey
  - Novartis Investigative Site, Lodi, New Jersey
  - Novartis Investigative Site, New Brunswick, New Jersey
  - Novartis Investigative Site, Ocean City, New Jersey
  - Novartis Investigative Site, Pomona, New Jersey
  - Novartis Investigative Site, Ridgewood, New Jersey
  - Novartis Investigative Site, Westwood, New Jersey
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Binghamton, New York
  - Novartis Investigative Site, Endwell, New York
  - Novartis Investigative Site, Kew Gardens, New York
  - Novartis Investigative Site, Mineola, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Rochester, New York
  - Novartis Investigative Site, Asheboro, North Carolina
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, Greenville, North Carolina
  - Novartis Investigative Site, Hickory, North Carolina
  - Novartis Investigative Site, Mooresville, North Carolina
  - Novartis Investigative Site, Pinehurst, North Carolina
  - Novartis Investigative Site, Salisbury, North Carolina
  - Novartis Investigative Site, Sanford, North Carolina
  - Novartis Investigative Site, Statesville, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Fargo, North Dakota
  - Novartis Investigative Site, Grand Forks, North Dakota
  - Novartis Investigative Site, Akron, Ohio
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Dayton, Ohio
  - Novartis Investigative Site, Marion, Ohio
  - Novartis Investigative Site, Bartlesville, Oklahoma
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Bend, Oregon
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Abington, Pennsylvania
  - Novartis Investigative Site, Altoona, Pennsylvania
  - Novartis Investigative Site, Beaver, Pennsylvania
  - Novartis Investigative Site, Bridgeville, Pennsylvania
  - Novartis Investigative Site, Camp Hill, Pennsylvania
  - Novartis Investigative Site, Erie, Pennsylvania
  - Novartis Investigative Site, Hershey, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Pottstown, Pennsylvania
  - Novartis Investigative Site, Uniontown, Pennsylvania
  - Novartis Investigative Site, Cumberland, Rhode Island
  - Novartis Investigative Site, Providence, Rhode Island
  - Novartis Investigative Site, Anderson, South Carolina
  - Novartis Investigative Site, Columbia, South Carolina
  - Novartis Investigative Site, Fort Mill, South Carolina
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Greer, South Carolina
  - Novartis Investigative Site, Moncks Corner, South Carolina
  - Novartis Investigative Site, Mt. Pleasant, South Carolina
  - Novartis Investigative Site, North Myrtle Beach, South Carolina
  - Novartis Investigative Site, Orangeburg, South Carolina
  - Novartis Investigative Site, Varnville, South Carolina
  - Novartis Investigative Site, Rapid City, South Dakota
  - Novartis Investigative Site, Sioux Falls, South Dakota
  - Novartis Investigative Site, Germantown, Tennessee
  - Novartis Investigative Site, Greenville, Tennessee
  - Novartis Investigative Site, Jackson, Tennessee
  - Novartis Investigative Site, Johnson City, Tennessee
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Allen, Texas
  - Novartis Investigative Site, Beaumont, Texas
  - Novartis Investigative Site, Bedford, Texas
  - Novartis Investigative Site, Brownsville, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Gonzales, Texas
  - Novartis Investigative Site, Greenville, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Irving, Texas
  - Novartis Investigative Site, Lake Jackson, Texas
  - Novartis Investigative Site, Leander, Texas
  - Novartis Investigative Site, Livingston, Texas
  - Novartis Investigative Site, Lufkin, Texas
  - Novartis Investigative Site, Marshall, Texas
  - Novartis Investigative Site, McAllen, Texas
  - Novartis Investigative Site, McKinney, Texas
  - Novartis Investigative Site, Odessa, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Sugar Land, Texas
  - Novartis Investigative Site, Temple, Texas
  - Novartis Investigative Site, Tomball, Texas
  - Novartis Investigative Site, Waco, Texas
  - Novartis Investigative Site, Webster, Texas
  - Novartis Investigative Site, Bountiful, Utah
  - Novartis Investigative Site, Layton, Utah
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Burke, Virginia
  - Novartis Investigative Site, Danville, Virginia
  - Novartis Investigative Site, Hopewell, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Port Orchard, Washington
  - Novartis Investigative Site, Renton, Washington
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Tacoma, Washington
  - Novartis Investigative Site, Madison, Wisconsin
- Argentina (24):
  - Novartis Investigative Site, Bahía Blanca, Buenos Aires
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Quilmes, Buenos Aires
  - Novartis Investigative Site, Ramos Mejía, Buenos Aires
  - Novartis Investigative Site, San Isidro, Buenos Aires
  - Novartis Investigative Site, San Nicolás de los Arroyos, Buenos Aires
  - Novartis Investigative Site, Zárate, Buenos Aires
  - Novartis Investigative Site, CABA, Buenos Aires F.D.
  - Novartis Investigative Site, San Salvador de Jujuy, Jujuy Province
  - Novartis Investigative Site, Posadas, Misiones Province
  - Novartis Investigative Site, Cipolletti, Río Negro Province
  - Novartis Investigative Site, San Miguel de Tucumán, San Miguel de Tucuman
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, CABA
  - Novartis Investigative Site, Corrientes
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Formosa
  - Novartis Investigative Site, Salta
  - Novartis Investigative Site, San Luis
  - Novartis Investigative Site, San Miguel de Tucumán
  - Novartis Investigative Site, Santa Fe
  - Novartis Investigative Site, Santiago del Estero
- Australia (12):
  - Novartis Investigative Site, Garran, Australian Capital Territory
  - Novartis Investigative Site, Gosford, New South Wales
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Liverpool, New South Wales
  - Novartis Investigative Site, Milton, Queensland
  - Novartis Investigative Site, Southport, Queensland
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, Bundoora, Victoria
  - Novartis Investigative Site, Geelong, Victoria
  - Novartis Investigative Site, Bateman, Western Australia
  - Novartis Investigative Site, Joondalup, Western Australia
  - Novartis Investigative Site, Perth, Western Australia
- Austria (5):
  - Novartis Investigative Site, Saint Stefan, Austria
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (13):
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Bonheiden
  - Novartis Investigative Site, Brasschaat
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, De Pinte
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Hasselt
  - Novartis Investigative Site, Huy
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Mechelen
  - Novartis Investigative Site, Ottignies
  - Novartis Investigative Site, Tienen
- Brazil (20):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Brasília, Federal District
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, Campo Grande, Mato Grosso do Sul
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Uberlândia, Minas Gerais
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Belém, Pará
  - Novartis Investigative Site, Recife, Pernambuco
  - Novartis Investigative Site, Passo Fundo, Rio Grande do Sul
  - Novartis Investigative Site, Pelotas, Rio Grande do Sul
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Blumenau, Santa Catarina
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, Santo André, São Paulo
  - Novartis Investigative Site, São José do Rio Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Tatuí, São Paulo
  - Novartis Investigative Site, Votuporanga, São Paulo
- Bulgaria (4):
  - Novartis Investigative Site, Pazardzhik
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
- Canada (33):
  - Novartis Investigative Site, New Westminster, British Columbia
  - Novartis Investigative Site, Surrey, British Columbia
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Mount Pearl, Newfoundland and Labrador
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Cambridge, Ontario
  - Novartis Investigative Site, Etobicoke, Ontario
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Kitchener, Ontario
  - Novartis Investigative Site, Mississauga, Ontario
  - Novartis Investigative Site, Newmarket, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Peterborough, Ontario
  - Novartis Investigative Site, Scarborough Village, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Drummondville, Quebec
  - Novartis Investigative Site, Gatineau, Quebec
  - Novartis Investigative Site, Granby, Quebec
  - Novartis Investigative Site, Joliette, Quebec
  - Novartis Investigative Site, Lachine, Quebec
  - Novartis Investigative Site, Laval, Quebec
  - Novartis Investigative Site, Lévis, Quebec
  - Novartis Investigative Site, Longueuil, Quebec
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
  - Novartis Investigative Site, Saint-Jean-sur-Richelieu, Quebec
  - Novartis Investigative Site, Sainte-Foy, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
  - Novartis Investigative Site, Ste-Foy, Quebec
  - Novartis Investigative Site, Terrebonne, Quebec
  - Novartis Investigative Site, Thetford-Mines, Quebec
  - Novartis Investigative Site, Saskatoon, Saskatchewan
- China (21):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Fuzhou, Fujian
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Nanning, Guangxi
  - Novartis Investigative Site, Shijiazhuang, Hebei
  - Novartis Investigative Site, Harbin, Heilongjiang
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Baotou, Inner Mongolia
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Colombia (13):
  - Novartis Investigative Site, Baranquilla, Atlántico
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Manizales, Caldas Department
  - Novartis Investigative Site, Cartegena, Colombia
  - Novartis Investigative Site, Cartagena, Departamento de Bolívar
  - Novartis Investigative Site, Bucaramanga, Santander Department
  - Novartis Investigative Site, Floridablanca, Santander Department
  - Novartis Investigative Site, Armenia
  - Novartis Investigative Site, Baranquilla
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Cali
  - Novartis Investigative Site, Florida Blanca
- Croatia (8):
  - Novartis Investigative Site, Varaždin, HRV
  - Novartis Investigative Site, Čakovec
  - Novartis Investigative Site, Koprivnica
  - Novartis Investigative Site, Krapinske Toplice
  - Novartis Investigative Site, Opatija
  - Novartis Investigative Site, Rijeka
  - Novartis Investigative Site, Virovitica
  - Novartis Investigative Site, Zagreb
- Czechia (30):
  - Novartis Investigative Site, Brandýs nad Labem, Czech Republic
  - Novartis Investigative Site, Jablonec nad Nisou, Czech Republic
  - Novartis Investigative Site, Kladno, Czech Republic
  - Novartis Investigative Site, Liberec, Czech Republic
  - Novartis Investigative Site, Louny, Czech Republic
  - Novartis Investigative Site, Ostrava, Czech Republic
  - Novartis Investigative Site, Pilsen, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Rožnov pod Radhoštěm, Czech Republic
  - Novartis Investigative Site, Semily, Czech Republic
  - Novartis Investigative Site, Svitavy, Czech Republic
  - Novartis Investigative Site, Třebíč, Czech Republic
  - Novartis Investigative Site, Ústí nad Labem, Czech Republic
  - Novartis Investigative Site, Ústí nad Orlicí, Czech Republic
  - Novartis Investigative Site, Vyškov, Czech Republic
  - Novartis Investigative Site, Znojmo, Czech Republic
  - Novartis Investigative Site, Most, CZE
  - Novartis Investigative Site, Prague, CZE
  - Novartis Investigative Site, Trutnov, CZE
  - Novartis Investigative Site, Benešov
  - Novartis Investigative Site, Brno-Bohunice
  - Novartis Investigative Site, Broumov
  - Novartis Investigative Site, Kolín
  - Novartis Investigative Site, Mariánské Lázně
  - Novartis Investigative Site, Pardubice
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Prague 4 - Krc
  - Novartis Investigative Site, Slaný
  - Novartis Investigative Site, Teplice
  - Novartis Investigative Site, Uherské Hradiště
- Estonia (6):
  - Novartis Investigative Site, Pärnu
  - Novartis Investigative Site, Saku
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
  - Novartis Investigative Site, Viljandi County
  - Novartis Investigative Site, Võru
- Germany (63):
  - Novartis Investigative Site, Muehlheim An Der Ruhr, North Rhine-Westphalia
  - Novartis Investigative Site, Bad Krozingen
  - Novartis Investigative Site, Balve
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Borna
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dillingen
  - Novartis Investigative Site, Dinslaken
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Duisburg
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Ebersbach
  - Novartis Investigative Site, Elsterwerda
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Falkensee
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Frankfurt am Main
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Fulda
  - Novartis Investigative Site, Giengen an der Brenz
  - Novartis Investigative Site, Görlitz
  - Novartis Investigative Site, Haag
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Heilbronn
  - Novartis Investigative Site, Huy / OT Anderbeck
  - Novartis Investigative Site, Jerichow
  - Novartis Investigative Site, Kallstadt
  - Novartis Investigative Site, Kamp-Lintfort
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Koblenz
  - Novartis Investigative Site, Künzing
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Lüneburg
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mayen
  - Novartis Investigative Site, Meissen
  - Novartis Investigative Site, Meißen
  - Novartis Investigative Site, Muehldorf Am Inn
  - Novartis Investigative Site, Mühlhausen
  - Novartis Investigative Site, Neuhofen
  - Novartis Investigative Site, Neunkirchen
  - Novartis Investigative Site, Northeim
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Oelde
  - Novartis Investigative Site, Oschatz
  - Novartis Investigative Site, Paderborn
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Rednitzhembach
  - Novartis Investigative Site, Reinfeld
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Rüdersdorf
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Wolmirstedt
- Greece (9):
  - Novartis Investigative Site, Crete Heraklion, Greece
  - Novartis Investigative Site, Heraklion Crete, Greece
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Magoula, GR
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Voula, GR
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Chalcis
  - Novartis Investigative Site, Pátrai
- Novartis Investigative Site, Guatemala City, Guatemala
- Hungary (14):
  - Novartis Investigative Site, Zalaegerszeg, Zala County
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Csongrád
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Gyula
  - Novartis Investigative Site, Kistarcsa
  - Novartis Investigative Site, Komárom
  - Novartis Investigative Site, Miskolc
  - Novartis Investigative Site, Mosonmagyaróvár
  - Novartis Investigative Site, Nyiregyháza
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Szentes
  - Novartis Investigative Site, Székesfehérvár
- Iceland (2):
  - Novartis Investigative Site, Kopavogur
  - Novartis Investigative Site, Reykjavik
- India (32):
  - Novartis Investigative Site, Hyderabad, Andhra Pradesh
  - Novartis Investigative Site, Nampally, Andhra Pradesh
  - Novartis Investigative Site, Nellore, Andhra Pradesh
  - Novartis Investigative Site, Tirupati, Andhra Pradesh
  - Novartis Investigative Site, Vijayawada, Andhra Pradesh
  - Novartis Investigative Site, Visakhapatnam, Andhra Pradesh
  - Novartis Investigative Site, Guntur, Andhrapradesh
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Surat, Gujarat
  - Novartis Investigative Site, Vadodara, Gujarat
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Bengaluru, Karnataka
  - Novartis Investigative Site, Manipal, Karnataka
  - Novartis Investigative Site, Kochi, Kerala
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Pune, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Ludhiana, Punjab
  - Novartis Investigative Site, Mohali, Punjab
  - Novartis Investigative Site, Bikaner, Rajasthan
  - Novartis Investigative Site, Jaipur, Rajasthan
  - Novartis Investigative Site, Rajasthan, Rajasthan
  - Novartis Investigative Site, Chennai, Tamil Nadu
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Madurai, Tamil Nadu
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Secunderabad, Telangana
  - Novartis Investigative Site, Ghaziabad, Uttar Pradesh
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
  - Novartis Investigative Site, Varanasi, Uttar Pradesh
  - Novartis Investigative Site, Ahmedabad
- Italy (33):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Fermo, AP
  - Novartis Investigative Site, Cortona, AR
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Treviglio, BG
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Montichiari, BS
  - Novartis Investigative Site, Monserrato, CA
  - Novartis Investigative Site, Santa Maria Capua Vetere, CE
  - Novartis Investigative Site, Chieti, CH
  - Novartis Investigative Site, Catanzaro, CZ
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Foggia, FG
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Pozzilli, IS
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Massa, MS
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Piacenza, PC
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Casorate Primo, PV
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Sassari, SS
  - Novartis Investigative Site, Palmanova, UD
  - Novartis Investigative Site, San Daniele del Friuli, UD
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Soriano Calabro, VV
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Novara
  - Novartis Investigative Site, Veruno
- Japan (36):
  - Novartis Investigative Site, Ichinomiya, Aichi-ken
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Seto, Aichi-ken
  - Novartis Investigative Site, Funabashi, Chiba
  - Novartis Investigative Site, Matsudo, Chiba
  - Novartis Investigative Site, Kasuga, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Onga-gun, Fukuoka
  - Novartis Investigative Site, Yukuhashi, Fukuoka
  - Novartis Investigative Site, Ōgaki, Gifu
  - Novartis Investigative Site, Fujioka, Gunma
  - Novartis Investigative Site, Takasaki, Gunma
  - Novartis Investigative Site, Hatsukaichi, Hiroshima
  - Novartis Investigative Site, Amagasaki, Hyōgo
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Takarazuka, Hyōgo
  - Novartis Investigative Site, Higashiibaraki-gun, Ibaraki
  - Novartis Investigative Site, Hitachi, Ibaraki
  - Novartis Investigative Site, Sakaidechō, Kagawa-ken
  - Novartis Investigative Site, Takamatsu, Kagawa-ken
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Nagano, Nagano
  - Novartis Investigative Site, Hirakata, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Sayama, Saitama
  - Novartis Investigative Site, Tokorozawa, Saitama
  - Novartis Investigative Site, Kusatsu, Shiga
  - Novartis Investigative Site, Komatsushimachō, Tokushima
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Fuchū, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
- Latvia (6):
  - Novartis Investigative Site, Liepāja, LV
  - Novartis Investigative Site, Riga, LV
  - Novartis Investigative Site, Ventspils, LV
  - Novartis Investigative Site, Daugavpils
  - Novartis Investigative Site, Riga
  - Novartis Investigative Site, Valmiera
- Lithuania (8):
  - Novartis Investigative Site, Kaunas, LTU
  - Novartis Investigative Site, Klaipėda, LTU
  - Novartis Investigative Site, Alytus
  - Novartis Investigative Site, Kaunas
  - Novartis Investigative Site, Kėdainiai
  - Novartis Investigative Site, Panevezys
  - Novartis Investigative Site, Šiauliai
  - Novartis Investigative Site, Vilnius
- Mexico (6):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, San Luis Potosí City, San Luis Potosí
  - Novartis Investigative Site, Culiacán, Sinaloa
  - Novartis Investigative Site, Aguascalientes
  - Novartis Investigative Site, Querétaro
  - Novartis Investigative Site, San Luis Potosí City
- Netherlands (23):
  - Novartis Investigative Site, Maastricht, AZ
  - Novartis Investigative Site, Apeldoorn, DZ
  - Novartis Investigative Site, Sneek, The Netherlands
  - Novartis Investigative Site, Alkmaar
  - Novartis Investigative Site, Amersfoort
  - Novartis Investigative Site, Amstelveen
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Breda
  - Novartis Investigative Site, Deventer
  - Novartis Investigative Site, Doetinchem
  - Novartis Investigative Site, Ede
  - Novartis Investigative Site, Gouda
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Haarlem
  - Novartis Investigative Site, Heerlen
  - Novartis Investigative Site, Hoorn
  - Novartis Investigative Site, Leeuwarden
  - Novartis Investigative Site, Meppel
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Tiel
  - Novartis Investigative Site, Utrecht
  - Novartis Investigative Site, Venlo
- Norway (15):
  - Novartis Investigative Site, Ålesund
  - Novartis Investigative Site, Elverum
  - Novartis Investigative Site, Hamar
  - Novartis Investigative Site, Harstad
  - Novartis Investigative Site, Hønefoss
  - Novartis Investigative Site, Lillehammer
  - Novartis Investigative Site, Moss
  - Novartis Investigative Site, Nesttun
  - Novartis Investigative Site, Oslo
  - Novartis Investigative Site, Sandefjord
  - Novartis Investigative Site, Skedsmokorset
  - Novartis Investigative Site, Stavanger
  - Novartis Investigative Site, Trondheim
  - Novartis Investigative Site, Tynset
  - Novartis Investigative Site, Tønsberg
- Peru (4):
  - Novartis Investigative Site, Bellavista, Lima region
  - Novartis Investigative Site, San Isidro, Lima region
  - Novartis Investigative Site, San Martín de Porres, Lima region
  - Novartis Investigative Site, Lima
- Poland (13):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Gdynia
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Ostrów Wielkopolski
  - Novartis Investigative Site, Oława
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Puławy
  - Novartis Investigative Site, Rumia
  - Novartis Investigative Site, Skierniewice
  - Novartis Investigative Site, Torun
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Węgrów
  - Novartis Investigative Site, Włocławek
- Puerto Rico (4):
  - Novartis Investigative Site, Manatí
  - Novartis Investigative Site, Mayagüez
  - Novartis Investigative Site, Ponce
  - Novartis Investigative Site, San Juan
- Romania (25):
  - Novartis Investigative Site, Piteşti, Argeş
  - Novartis Investigative Site, Bucharest, District 1
  - Novartis Investigative Site, Bucharest, District 2
  - Novartis Investigative Site, Bucharest, District 4
  - Novartis Investigative Site, Oradea, Jud Bihor
  - Novartis Investigative Site, Cluj-Napoca, Jud Cluj
  - Novartis Investigative Site, Iași, Jud Iasi
  - Novartis Investigative Site, Târgu Mureş, Jud Mures
  - Novartis Investigative Site, Constanța, Jud. Constanta
  - Novartis Investigative Site, Craiova, Jud. Dolj
  - Novartis Investigative Site, Iași, Jud. Iasi
  - Novartis Investigative Site, Târgu Mureş, Mureș County
  - Novartis Investigative Site, Tg Mures, Mureș County
  - Novartis Investigative Site, Brăila, ROM
  - Novartis Investigative Site, Timișoara, Timiș County
  - Novartis Investigative Site, Baia Mare
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Bucharest
  - Novartis Investigative Site, Cluj-Napoca
  - Novartis Investigative Site, Craiova
  - Novartis Investigative Site, Oradea
  - Novartis Investigative Site, Piteşti
  - Novartis Investigative Site, Sibiu
  - Novartis Investigative Site, Târgu Mureş
  - Novartis Investigative Site, Timișoara
- Russia (23):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Izhevsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Kirov
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Novosibirsk
  - Novartis Investigative Site, Penza
  - Novartis Investigative Site, Perm
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Samara
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Sestroretsk
  - Novartis Investigative Site, Smolensk
  - Novartis Investigative Site, Syktyvkar
  - Novartis Investigative Site, Tomsk
  - Novartis Investigative Site, Tyumen
  - Novartis Investigative Site, Vladimir
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Serbia (4):
  - Novartis Investigative Site, Belgrade
  - Novartis Investigative Site, Kamenitz
  - Novartis Investigative Site, Niš
  - Novartis Investigative Site, Niška Banja
- Slovakia (24):
  - Novartis Investigative Site, Bratislava, Slovak Republic
  - Novartis Investigative Site, Brezno, Slovak Republic
  - Novartis Investigative Site, Komárno, Slovak Republic
  - Novartis Investigative Site, Košice, Slovak Republic
  - Novartis Investigative Site, Považská Bystrica, Slovak Republic
  - Novartis Investigative Site, Prešov, Slovak Republic
  - Novartis Investigative Site, Rimavská Sobota, Slovak Republic
  - Novartis Investigative Site, Svidník, Slovak Republic
  - Novartis Investigative Site, Veľký Krtíš, Slovak Republic
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Bardejov
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Dubnica nad Váhom
  - Novartis Investigative Site, Dunajská Streda
  - Novartis Investigative Site, Galanta
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Levice
  - Novartis Investigative Site, Lučenec
  - Novartis Investigative Site, Martin
  - Novartis Investigative Site, Nitra
  - Novartis Investigative Site, Nové Zámky
  - Novartis Investigative Site, Prešov
  - Novartis Investigative Site, Trnava
  - Novartis Investigative Site, Žilina
- Slovenia (3):
  - Novartis Investigative Site, Celje
  - Novartis Investigative Site, Golnik
  - Novartis Investigative Site, Ljubljana
- South Africa (10):
  - Novartis Investigative Site, Durban, KwaZulu-Natal
  - Novartis Investigative Site, Cape Town, Western Cape
  - Novartis Investigative Site, Alberton
  - Novartis Investigative Site, Bloemfontein
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Centurion
  - Novartis Investigative Site, Johannesburg
  - Novartis Investigative Site, Kempton Park
  - Novartis Investigative Site, Pretoria
  - Novartis Investigative Site, Western Cape
- South Korea (10):
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Uijeongbu-si, Gyeonggi-do
  - Novartis Investigative Site, Daejeon, Korea
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Daegu
  - Novartis Investigative Site, Gwangju
  - Novartis Investigative Site, Seoul
- Sweden (15):
  - Novartis Investigative Site, Gothenburg, Västra Götaland County
  - Novartis Investigative Site, Borås
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Kristianstad
  - Novartis Investigative Site, Luleå
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Malmo
  - Novartis Investigative Site, Mölndal
  - Novartis Investigative Site, Östersund
  - Novartis Investigative Site, Skanör
  - Novartis Investigative Site, Skellefteå
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uddevalla
  - Novartis Investigative Site, Vällingby
  - Novartis Investigative Site, Västerås
- Taiwan (9):
  - Novartis Investigative Site, Taichung, Taiwan ROC
  - Novartis Investigative Site, Taipei, Taiwan, ROC
  - Novartis Investigative Site, Changhua
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
  - Novartis Investigative Site, Yilan
- Turkey (Türkiye) (7):
  - Novartis Investigative Site, Eskişehir, Meselik
  - Novartis Investigative Site, Aydin
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Mersin
  - Novartis Investigative Site, Sivas
- United Kingdom (30):
  - Novartis Investigative Site, Basingstoke, Hampshire
  - Novartis Investigative Site, Newport, Isle Of Wight
  - Novartis Investigative Site, Salford, Manchester
  - Novartis Investigative Site, Whitby, North Yorkshire
  - Novartis Investigative Site, Dundee, Perthshire
  - Novartis Investigative Site, Axbridge, Somerset
  - Novartis Investigative Site, Taunton, Somerset
  - Novartis Investigative Site, Cardiff, Wales
  - Novartis Investigative Site, Barnet
  - Novartis Investigative Site, Berkshire
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Cheshire
  - Novartis Investigative Site, Chesterfield
  - Novartis Investigative Site, Chorley
  - Novartis Investigative Site, Exeter
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Irvine
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Newport
  - Novartis Investigative Site, Norwich
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Sheffield
  - Novartis Investigative Site, Wiltshire
  - Novartis Investigative Site, Worcester
  - Novartis Investigative Site, York

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Woo J, Lu D, Lewandowski A, Xu H, Serrano P, Healey M, Yates DP, Beste MT, Libby P, Ridker PM, Steensma DP. Effects of IL-1beta inhibition on anemia and clonal hematopoiesis in the randomized CANTOS trial. Blood Adv. 2023 Dec 26;7(24):7471-7484. doi: 10.1182/bloodadvances.2023011578. PMID 37934948
- [Derived] Ridker PM, Tuttle KR, Perkovic V, Libby P, MacFadyen JG. Inflammation drives residual risk in chronic kidney disease: a CANTOS substudy. Eur Heart J. 2022 Dec 7;43(46):4832-4844. doi: 10.1093/eurheartj/ehac444. PMID 35943897
- [Derived] Svensson EC, Madar A, Campbell CD, He Y, Sultan M, Healey ML, Xu H, D'Aco K, Fernandez A, Wache-Mainier C, Libby P, Ridker PM, Beste MT, Basson CT. TET2-Driven Clonal Hematopoiesis and Response to Canakinumab: An Exploratory Analysis of the CANTOS Randomized Clinical Trial. JAMA Cardiol. 2022 May 1;7(5):521-528. doi: 10.1001/jamacardio.2022.0386. PMID 35385050
- [Derived] Everett BM, MacFadyen JG, Thuren T, Libby P, Glynn RJ, Ridker PM. Inhibition of Interleukin-1beta and Reduction in Atherothrombotic Cardiovascular Events in the CANTOS Trial. J Am Coll Cardiol. 2020 Oct 6;76(14):1660-1670. doi: 10.1016/j.jacc.2020.08.011. PMID 33004131
- [Derived] Schieker M, Conaghan PG, Mindeholm L, Praestgaard J, Solomon DH, Scotti C, Gram H, Thuren T, Roubenoff R, Ridker PM. Effects of Interleukin-1beta Inhibition on Incident Hip and Knee Replacement : Exploratory Analyses From a Randomized, Double-Blind, Placebo-Controlled Trial. Ann Intern Med. 2020 Oct 6;173(7):509-515. doi: 10.7326/M20-0527. Epub 2020 Aug 4. PMID 32744862
- [Derived] Vallurupalli M, MacFadyen JG, Glynn RJ, Thuren T, Libby P, Berliner N, Ridker PM. Effects of Interleukin-1beta Inhibition on Incident Anemia: Exploratory Analyses From a Randomized Trial. Ann Intern Med. 2020 Apr 21;172(8):523-532. doi: 10.7326/M19-2945. Epub 2020 Mar 24. PMID 32203978
- [Derived] Rothman AM, MacFadyen J, Thuren T, Webb A, Harrison DG, Guzik TJ, Libby P, Glynn RJ, Ridker PM. Effects of Interleukin-1beta Inhibition on Blood Pressure, Incident Hypertension, and Residual Inflammatory Risk: A Secondary Analysis of CANTOS. Hypertension. 2020 Feb;75(2):477-482. doi: 10.1161/HYPERTENSIONAHA.119.13642. Epub 2019 Dec 30. PMID 31884854
- [Derived] Ridker PM, MacFadyen JG, Thuren T, Libby P. Residual inflammatory risk associated with interleukin-18 and interleukin-6 after successful interleukin-1beta inhibition with canakinumab: further rationale for the development of targeted anti-cytokine therapies for the treatment of atherothrombosis. Eur Heart J. 2020 Jun 14;41(23):2153-2163. doi: 10.1093/eurheartj/ehz542. PMID 31504417
- [Derived] Everett BM, Cornel JH, Lainscak M, Anker SD, Abbate A, Thuren T, Libby P, Glynn RJ, Ridker PM. Anti-Inflammatory Therapy With Canakinumab for the Prevention of Hospitalization for Heart Failure. Circulation. 2019 Mar 5;139(10):1289-1299. doi: 10.1161/CIRCULATIONAHA.118.038010. PMID 30586730
- [Derived] Solomon DH, Glynn RJ, MacFadyen JG, Libby P, Thuren T, Everett BM, Ridker PM. Relationship of Interleukin-1beta Blockade With Incident Gout and Serum Uric Acid Levels: Exploratory Analysis of a Randomized Controlled Trial. Ann Intern Med. 2018 Oct 16;169(8):535-542. doi: 10.7326/M18-1167. Epub 2018 Sep 18. PMID 30242335
- [Derived] Ridker PM, Libby P, MacFadyen JG, Thuren T, Ballantyne C, Fonseca F, Koenig W, Shimokawa H, Everett BM, Glynn RJ. Modulation of the interleukin-6 signalling pathway and incidence rates of atherosclerotic events and all-cause mortality: analyses from the Canakinumab Anti-Inflammatory Thrombosis Outcomes Study (CANTOS). Eur Heart J. 2018 Oct 7;39(38):3499-3507. doi: 10.1093/eurheartj/ehy310. PMID 30165610
- [Derived] Ridker PM, MacFadyen JG, Glynn RJ, Koenig W, Libby P, Everett BM, Lefkowitz M, Thuren T, Cornel JH. Inhibition of Interleukin-1beta by Canakinumab and Cardiovascular Outcomes in Patients With Chronic Kidney Disease. J Am Coll Cardiol. 2018 May 29;71(21):2405-2414. doi: 10.1016/j.jacc.2018.03.490. PMID 29793629
- [Derived] Everett BM, Donath MY, Pradhan AD, Thuren T, Pais P, Nicolau JC, Glynn RJ, Libby P, Ridker PM. Anti-Inflammatory Therapy With Canakinumab for the Prevention and Management of Diabetes. J Am Coll Cardiol. 2018 May 29;71(21):2392-2401. doi: 10.1016/j.jacc.2018.03.002. Epub 2018 Mar 12. PMID 29544870
- [Derived] Ridker PM, MacFadyen JG, Everett BM, Libby P, Thuren T, Glynn RJ; CANTOS Trial Group. Relationship of C-reactive protein reduction to cardiovascular event reduction following treatment with canakinumab: a secondary analysis from the CANTOS randomised controlled trial. Lancet. 2018 Jan 27;391(10118):319-328. doi: 10.1016/S0140-6736(17)32814-3. Epub 2017 Nov 13. PMID 29146124
- [Derived] Ridker PM, MacFadyen JG, Thuren T, Everett BM, Libby P, Glynn RJ; CANTOS Trial Group. Effect of interleukin-1beta inhibition with canakinumab on incident lung cancer in patients with atherosclerosis: exploratory results from a randomised, double-blind, placebo-controlled trial. Lancet. 2017 Oct 21;390(10105):1833-1842. doi: 10.1016/S0140-6736(17)32247-X. Epub 2017 Aug 27. PMID 28855077
- [Derived] Ridker PM, Everett BM, Thuren T, MacFadyen JG, Chang WH, Ballantyne C, Fonseca F, Nicolau J, Koenig W, Anker SD, Kastelein JJP, Cornel JH, Pais P, Pella D, Genest J, Cifkova R, Lorenzatti A, Forster T, Kobalava Z, Vida-Simiti L, Flather M, Shimokawa H, Ogawa H, Dellborg M, Rossi PRF, Troquay RPT, Libby P, Glynn RJ; CANTOS Trial Group. Antiinflammatory Therapy with Canakinumab for Atherosclerotic Disease. N Engl J Med. 2017 Sep 21;377(12):1119-1131. doi: 10.1056/NEJMoa1707914. Epub 2017 Aug 27. PMID 28845751
- [Derived] Canada JM, Fronk DT, Cei LF, Carbone S, Erdle CO, Abouzaki NA, Melchior RD, Thomas CS, Christopher S, Turlington JS, Trankle CR, Thurber CJ, Evans RK, Dixon DL, Van Tassell BW, Arena R, Abbate A. Usefulness of C-Reactive Protein Plasma Levels to Predict Exercise Intolerance in Patients With Chronic Systolic Heart Failure. Am J Cardiol. 2016 Jan 1;117(1):116-20. doi: 10.1016/j.amjcard.2015.10.020. Epub 2015 Oct 19. PMID 26546248
- [Derived] Ridker PM, Thuren T, Zalewski A, Libby P. Interleukin-1beta inhibition and the prevention of recurrent cardiovascular events: rationale and design of the Canakinumab Anti-inflammatory Thrombosis Outcomes Study (CANTOS). Am Heart J. 2011 Oct;162(4):597-605. doi: 10.1016/j.ahj.2011.06.012. Epub 2011 Sep 14. PMID 21982649

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10066 patients enrolled in the Core phase (4 randomized groups); 5 patients enrolled in the safety set were not included in efficacy set. 5777 patients continued in the Extension phase (539 entered only the washout period, 5238 entered the treatment period(s)). The Core phase completed as planned; "terminated" applies to the Extension phase.
Pre-assignment Details: A total of 17482 patients were screened, and 10102 patients completed the screening phase. A total of 6430 patients did not complete the screening phase due to screen failure.
Groups:
- Group I: Core phase: Blinded Canakinumab 300 mg quarterly subcutaneous + standard of care (SoC) therapy Extension phase: Switched to open-label Canakinumab 150 mg quarterly subcutaneous + standard of care (SoC) therapy
- Group II: Core phase: Blinded Canakinumab 150 mg quarterly subcutaneous + standard of care (SoC) therapy Extension phase: Switched to open-label Canakinumab 150 mg quarterly subcutaneous + standard of care (SoC) therapy
- Group III: Core phase: Blinded Canakinumab 50 mg quarterly subcutaneous + standard of care (SoC) therapy Extension phase: Switched to open-label Canakinumab 150 mg quarterly subcutaneous + standard of care (SoC) therapy
- Group IV: Core phase: Blinded matching placebo quarterly subcutaneous + standard of care (SoC) therapy Extension phase: Switched to open-label Canakinumab 150 mg quarterly subcutaneous + standard of care (SoC) therapy
Period: Core Phase
Arm/Group | Group I | Group II | Group III | Group IV
Started | 2263 | 2284 | 2170 | 3344
Completed | 2235 | 2252 | 2144 | 3311
Not Completed | 28 | 32 | 26 | 33
Not completed — Subject decision (vital status: missing) | 1 | 2 | 2 | 1
Not completed — Subject decision (vital stat: unkn) | 0 | 0 | 3 | 3
Not completed — Subject decision (vital stat: dead) | 1 | 3 | 4 | 4
Not completed — Subject decision (vital stat: alive) | 23 | 24 | 13 | 20
Not completed — Lost to Follow-up | 3 | 3 | 4 | 5
Period: Extension Phase
Arm/Group | Group I | Group II | Group III | Group IV
Started | 1267 | 1287 | 1279 | 1944
Stopped/Discontinued Study at Washout | 127 | 97 | 137 | 178
Completed Treatment Period | 41 | 45 | 49 | 60
Details Missing | 0 | 1 | 1 | 0
Completed | 168 | 143 | 187 | 238
Not Completed | 1099 | 1144 | 1092 | 1706
Not completed — Study terminated by sponsor | 1073 | 1124 | 1067 | 1660
Not completed — Withdrawal by Subject | 20 | 13 | 19 | 37
Not completed — Lost to Follow-up | 4 | 3 | 4 | 7
Not completed — Technical Problems | 2 | 4 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) - All randomized patients except for those who were misrandomized or from sites with serious GCP violations.
  Baseline characteristics data are presented for patients enrolled in the Core phase of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I | Group II | Group III | Group IV | Total
Number analyzed (Participants) | 2263 | 2284 | 2170 | 3344 | 10061
Age, Customized [Number; unit: Participants] — Population: FAS
  Participants
    < 65 | 1424 | 1428 | 1350 | 2089 | 6291
    >= 65 | 839 | 856 | 820 | 1255 | 3770
Sex: Female, Male [Count of Participants; unit: Participants] — Population: FAS
  Participants
    Female | 606 | 575 | 541 | 865 | 2587
    Male | 1657 | 1709 | 1629 | 2479 | 7474
Race/Ethnicity, Customized [Number; unit: Participants] — Population: FAS
  Participants
    Caucasian | 1804 | 1808 | 1772 | 2652 | 8036
    Black | 84 | 67 | 61 | 106 | 318
    Asian | 265 | 278 | 232 | 388 | 1163
    Native American | 47 | 49 | 41 | 82 | 219
    Pacific Islander | 0 | 0 | 1 | 1 | 2
    Unknown | 3 | 3 | 1 | 3 | 10
    Other | 60 | 79 | 62 | 112 | 313

OUTCOME MEASURES:

1. Primary Outcome: Analysis of Core Phase First CEC Confirmed Major Adverse Cardiovascular Events (MACE) and Its Components
Description: Time to occurrence of CEC (Cardiovascular clinical events adjudication committee) confirmed MACE, which was a composite endpoint consisting of CEC confirmed CV death, CEC confirmed non-fatal MI,or CEC confirmed non-fatal stroke. Patients with the CEC adjudicated reason for death of "Unknown" were counted as CV (cardiovascular) death.
Time Frame: From randomization, to end of treatment plus 30 days, up to approximately 6 years
Population: Full Analysis Set (FAS): All randomized patients except for those who were misrandomized or from sites with serious GCP violations
Measure: Number; unit: Participants
Arm/Group | Group I | Group II | Group III | Group IV
Number analyzed (Participants) | 2263 | 2284 | 2170 | 3344
Participants
  MACE | 322 | 320 | 313 | 535
  CV death | 151 | 144 | 137 | 235
  MI (fatal and non-fatal) | 174 | 159 | 169 | 292
  MI (non-fatal) | 171 | 158 | 168 | 291
  Stroke (fatal and non-fatal) | 51 | 63 | 58 | 92
  Stroke (non-fatal) | 51 | 63 | 58 | 91
Statistical Analysis 1: Comparison: Group I vs Group IV; H11: The hazard rate of first adjudication committee confirmed MACE in the canakinumab 300 mg dose group is greater than or equal to the hazard rate of the placebo group; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.0648, Log Rank — 1-sided adjusted for multiplicity using weighted Dunnett test. [significance level 0.0245]; Cox Proportional Hazard = 0.86, 95% CI 2-sided [0.75 to 0.99] — MACE
Statistical Analysis 2: Comparison: Group II vs Group IV; H21: The hazard rate of first adjudication committee confirmed MACE in the canakinumab 150 mg dose group is greater than or equal to the hazard rate of the placebo group; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.0241, Log Rank — 1-sided adjusted for multiplicity using weighted Dunnett test. [significance level 0.0245]; Cox Proportional Hazard = 0.85, 95% CI 2-sided [0.74 to 0.98] — MACE
Statistical Analysis 3: Comparison: Group III vs Group IV; H31: The hazard rate of first adjudication committee confirmed MACE in the canakinumab 50 mg dose group is greater than or equal to the hazard rate of the placebo group; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.1895, Log Rank — 1-sided adjusted for multiplicity using weighted Dunnett test. [significance level 0.0245]; Cox Proportional Hazard = 0.93, 95% CI 2-sided [0.80 to 1.07] — MACE
Statistical Analysis 4: Comparison: Group I vs Group IV; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.572, Regression, Cox — 2-sided unadjusted p-value; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.77 to 1.16] — CV death
Statistical Analysis 5: Comparison: Group II vs Group IV; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.296, Regression, Cox — 2-sided unadjusted p-value; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.73 to 1.10] — CV death
Statistical Analysis 6: Comparison: Group III vs Group IV; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.369, Regression, Cox — 2-sided unadjusted p-value; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.73 to 1.12] — CV death
Statistical Analysis 7: Comparison: Group I vs Group IV; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.067, Regression, Cox — 2-sided unadjusted p-value; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.69 to 1.01] — MI (fatal and non-fatal)
Statistical Analysis 8: Comparison: Group II vs Group IV; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.006, Regression, Cox — 2-sided unadjusted p-value; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.63 to 0.92] — MI (fatal and non-fatal)
Statistical Analysis 9: Comparison: Group III vs Group IV; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.542, Regression, Cox — 2-sided unadjusted p-value; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.78 to 1.14] — MI (fatal and non-fatal)
Statistical Analysis 10: Comparison: Group I vs Group IV; Test type: Other — A HR < 1 favors Canakinumab; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.68 to 1.00] — MI (non-fatal)
Statistical Analysis 11: Comparison: Group II vs Group IV; Test type: Other — A HR < 1 favors Canakinumab; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.62 to 0.92] — MI (non-fatal)
Statistical Analysis 12: Comparison: Group III vs Group IV; Test type: Other — A HR < 1 favors Canakinumab; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.78 to 1.14] — MI (non-fatal)
Statistical Analysis 13: Comparison: Group I vs Group IV; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.190, Regression, Cox — 2-sided unadjusted p-value; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.56 to 1.12] — Stroke (fatal and non-fatal)
Statistical Analysis 14: Comparison: Group II vs Group IV; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.912, Regression, Cox — 2-sided unadjusted p-value; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.71 to 1.35] — Stroke (fatal and non-fatal)
Statistical Analysis 15: Comparison: Group III vs Group IV; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.871, Regression, Cox — 2-sided unadjusted p-value; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.74 to 1.43] — Stroke (fatal and non-fatal)
Statistical Analysis 16: Comparison: Group I vs Group IV; Test type: Other — A HR < 1 favors Canakinumab; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.57 to 1.13] — Stroke (nonfatal)
Statistical Analysis 17: Comparison: Group II vs Group IV; Test type: Other — A HR < 1 favors Canakinumab; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.72 to 1.37] — Stroke (nonfatal)
Statistical Analysis 18: Comparison: Group III vs Group IV; Test type: Other — A HR < 1 favors Canakinumab; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.75 to 1.45] — Stroke (nonfatal)

2. Primary Outcome: Substudy 1 (Core Phase): Change From Baseline in Carotid Plaque Burden in the Bifurcation Region of the Index Carotid Artery
Time Frame: 24 months
Population: Data from subjects were not collected as the substudy was terminated prior to data collection.
Arm/Group | Group I | Group II | Group III | Group IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Primary Outcome: Substudy 2 (Core Phase): Change From Baseline of the Insulin Secretion Rate (ISR) Relative to Glucose 0-30 Min Defined as Φ30 = AUCISR 0-30 / AUCGluc 0-30 Averaged Across the Year 3, 4, 5 Visits
Time Frame: From randomization up to approximately 6 years
Population: Data from subjects were not collected as the substudy was terminated prior to data collection.
Arm/Group | Group I | Group II | Group III | Group IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Patients With Core Phase CEC Confirmed CV Death, Non-fatal MI, Non-fatal Stroke, or Hospitalization for Unstable Angina Requiring Unplanned Revascularization
Description: Occurrence of the composite cardiovascular endpoint consisting of cardiovascular death, non-fatal MI, non-fatal stroke or hospitalization for unstable angina requiring unplanned revascularization.
  MACE includes CV death, non-fatal MI and non-fatal stroke. CEC = Clinical Endpoints Committee
Time Frame: From randomization, to end of treatment pus 30 days, up to approximately 6 years
Population: FAS: All randomized patients except for those who were misrandomized or from sites with serious GCP violations
Measure: Number; unit: Participants
Arm/Group | Group I | Group II | Group III | Group IV
Number analyzed (Participants) | 2263 | 2284 | 2170 | 3344
Participants
  MACE or unstable angina | 348 | 352 | 344 | 601
  Unstable angina | 34 | 38 | 38 | 85
Statistical Analysis 1: Comparison: Group I vs Group IV; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.0648, Log Rank — 1-sided adjusted for multiplicity using weighted Dunnett test. [significance level 0.0245]; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.72 to 0.94] — MACE or unstable angina
Statistical Analysis 2: Comparison: Group II vs Group IV; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.0241, Log Rank — 1-sided adjusted for multiplicity using weighted Dunnett test. [significance level 0.0245]; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.73 to 0.95] — MACE or unstable angina
Statistical Analysis 3: Comparison: Group III vs Group IV; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.1895, Log Rank — 1-sided adjusted for multiplicity using weighted Dunnett test. [significance level 0.0245]; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.79 to 1.03] — MACE or unstable angina
Statistical Analysis 4: Comparison: Group I vs Group IV; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.007, Regression, Cox — 2-sided unadjusted p-value; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.39 to 0.86] — unstable angina
Statistical Analysis 5: Comparison: Group II vs Group IV; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.022, Regression, Cox — 2-sided unadjusted p-value; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.44 to 0.94] — unstable angina
Statistical Analysis 6: Comparison: Group III vs Group IV; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.086, Regression, Cox — 2-sided unadjusted p-value; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.48 to 1.05] — unstable angina

5. Secondary Outcome: Patients With Core Phase New Onset Type 2 Diabetes Among Patients With Pre-diabetes at Randomization
Description: Time to CEC confirmed new onset of type 2 diabetes among those with pre-diabetes at randomization (i.e. excluding those that are normoglycemic at baseline)
Time Frame: From randomization up to approximately 6 years
Population: FAS: All randomized patients except for those who were misrandomized or from sites with serious GCP violations
Measure: Number; unit: Participants
Arm/Group | Group I | Group II | Group III | Group IV
Number analyzed (Participants) | 1132 | 1094 | 1089 | 1645
Participants | 169 | 171 | 161 | 246
Statistical Analysis 1: Comparison: Group I vs Group IV; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.8456, Log Rank — 1-sided adjusted for multiplicity using weighted Dunnett test. [significance level 0.0245]; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.83 to 1.23]
Statistical Analysis 2: Comparison: Group II vs Group IV; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.8456, Log Rank — 1-sided adjusted for multiplicity using weighted Dunnett test. [significance level 0.0245]; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.87 to 1.29]
Statistical Analysis 3: Comparison: Group III vs Group IV; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.6541, Log Rank — 1-sided adjusted for multiplicity using weighted Dunnett test. [significance level 0.0245]; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.80 to 1.20]

6. Secondary Outcome: Core Phase All-cause Mortality, Non-fatal MI, or Non-fatal Stroke
Description: Occurrence of the composite endpoint consisting of all-cause mortality, non-fatal IM, or non-fatal stroke
Time Frame: From randomization, to end of treatment plus 30 days, up to approximately 6 years
Population: FAS: All randomized patients except for those who were misrandomized or from sites with serious GCP violations
Measure: Number; unit: Participants
Arm/Group | Group I | Group II | Group III | Group IV
Number analyzed (Participants) | 2263 | 2284 | 2170 | 3344
Participants | 403 | 395 | 394 | 661
Statistical Analysis 1: Comparison: Group I vs Group IV; Test type: Superiority; p = 0.028, Regression, Cox — 2-sided unadjusted p-value; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.77 to 0.99] — All-cause mortality or MI or Stroke
Statistical Analysis 2: Comparison: Group II vs Group IV; Test type: Superiority; p = 0.011, Regression, Cox — 2-sided unadjusted p-value; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.75 to 0.96] — All-cause mortality or MI or Stroke
Statistical Analysis 3: Comparison: Group III vs Group IV; Test type: Superiority; p = 0.377, Regression, Cox — 2-sided unadjusted p-value; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.83 to 1.07] — All-cause mortality or MI or Stroke

7. Secondary Outcome: Core Phase All-cause Mortality
Description: Number of participant deaths
Time Frame: From randomization, to end of treatment plus 30 days, up to approximately 6 years
Population: FAS: All randomized patients except for those who were misrandomized or from sites with serious GCP violations
Measure: Number; unit: Participants
Arm/Group | Group I | Group II | Group III | Group IV
Number analyzed (Participants) | 2263 | 2284 | 2170 | 3344
Participants | 239 | 238 | 228 | 375
Statistical Analysis 1: Comparison: Group I vs Group IV; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.406, Regression, Cox — 2-sided unadjusted p-value; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.79 to 1.10] — All-cause mortality
Statistical Analysis 2: Comparison: Group II vs Group IV; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.329, Regression, Cox — 2-sided unadjusted p-value; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.78 to 1.09] — All-cause mortality
Statistical Analysis 3: Comparison: Group III vs Group IV; Test type: Superiority — A HR < 1 favors Canakinumab; p = 0.597, Regression, Cox — 2-sided unadjusted p-value; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.81 to 1.13] — All-cause mortality

8. Secondary Outcome: Summary of Adverse Events (Core Phase)
Description: Summary of Adverse Events (AEs) and Serious Adverse Events (SAEs) occurring during the double-blind Core phase of the study. AEs/SAEs are any signs or symptoms that occur during the study treatment.
Time Frame: From randomization, to end of treatment plus 30 days, up to approximately 6 years
Population: Safety set: All patients who received at least one dose of study treatment and had at least one post-baseline safety assessment
Measure: Number; unit: Participants
Arm/Group | Group I | Group II | Group III | Group IV
Number analyzed (Participants) | 2263 | 2285 | 2170 | 3348
Participants
  Patients with at least one AE | 1987 | 1970 | 1872 | 2915
  AEs suspected to be related tostudy drug | 355 | 350 | 267 | 474
  Patients with at least one SAE | 836 | 812 | 741 | 1204
  Discontinued due to SAEs | 135 | 130 | 117 | 198
  Discontinued due to non-seriousAEs | 40 | 34 | 26 | 47
  AEs leading to study treatmentinterruption | 268 | 270 | 228 | 399

9. Secondary Outcome: Summary of Adverse Events (Extension Phase)
Description: Summary of Adverse Events (AEs) and Serious Adverse Events (SAEs) occurring during the Extension phase of the study. AEs/SAEs are any signs or symptoms that occur during the study treatment.
Time Frame: From start of Extension phase, to end of treatment plus 30 days, up to approximately 2 years
Population: Extension Safety set: All patients who received at least one dose of study treatment during the Core Phase and who entered the Extension phase.
Measure: Number; unit: Participants
Arm/Group | Group I | Group II | Group III | Group IV
Number analyzed (Participants) | 1267 | 1287 | 1279 | 1944
Participants
  Patients with at least one AE | 788 | 845 | 793 | 1250
  AEs suspected to be related tostudy drug | 40 | 34 | 43 | 65
  Patients with at least one SAE | 310 | 326 | 322 | 465
  Discontinued due to SAEs | 67 | 71 | 71 | 98
  Discontinued due to non-seriousAEs | 8 | 6 | 12 | 8
  AEs leading to study treatmentinterruption | 59 | 72 | 62 | 100

10. Secondary Outcome: Substudy 1 (Core Phase): Change From Baseline of the Total Vessel Wall Area at Month 3 in the Bifurcation Region of the Index Carotid Artery
Time Frame: 3 months
Population: Data from subjects were not collected as the substudy was terminated prior to data collection.
Arm/Group | Group I | Group II | Group III | Group IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Substudy 1 (Core Phase): Mean Total Vessel Wall Area Across the Left and Right Carotid Artery at Month 3 and Month 24
Time Frame: 24 months
Population: Data from subjects were not collected as the substudy was terminated prior to data collection.
Arm/Group | Group I | Group II | Group III | Group IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Substudy 1 (Core Phase): Change From Baseline in Corresponding Total Vessel Wall Area in the Left and Right Carotid Arteries
Time Frame: 24 months
Population: Data from subjects were not collected as the substudy was terminated prior to data collection.
Arm/Group | Group I | Group II | Group III | Group IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Substudy 1 (Core Phase): The Existence of a Baseline Total Vessel Wall Area by Treatment Interaction as Well as the Consistency of the Treatment Effect Across Subgroups
Time Frame: 24 months
Population: Data from subjects were not collected as the substudy was terminated prior to data collection.
Arm/Group | Group I | Group II | Group III | Group IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Substudy 2 (Core Phase): Change From Baseline in Insulin Sensitivity Index
Time Frame: From randomization up to approximately 6 years
Population: Data from subjects were not collected as the substudy was terminated prior to data collection.
Arm/Group | Group I | Group II | Group III | Group IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Substudy 2 (Core Phase): Change From Baseline in OGTT Stimulated Area Under Curve (AUC) 0-120 Min of Glucose Concentration, Insulin Concentration, Pro-insulin Concentration, and Insulin Concentration/Glucose Concentration Ratio
Time Frame: From randomization up to approximately 6 years
Population: Data from subjects were not collected as the substudy was terminated prior to data collection.
Arm/Group | Group I | Group II | Group III | Group IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Secondary Outcome: Substudy 2 (Core Phase): Change From Baseline in Fasting Pro-Insulin Concentration/Insulin Concentration Ratio
Time Frame: From randomization up to approximately 6 years
Population: Data from subjects were not collected as the substudy was terminated prior to data collection.
Arm/Group | Group I | Group II | Group III | Group IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

17. Secondary Outcome: Substudy 2 (Core Phase): Change From Baseline in OGTT Stimulated Area Under the Curve (AUC) 0-120 Min of C-peptide Concentration
Time Frame: From randomization up to approximately 6 years
Population: Data from subjects were not collected as the substudy was terminated prior to data collection.
Arm/Group | Group I | Group II | Group III | Group IV
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Core phase: From randomization to end of treatment plus 30 days; up to approximately 6 years; Extension phase: From start of Extension phase, to end of treatment plus 30 days, up to approximately 2 years.
Description: AEs/SAEs are any signs or symptoms that occur during the study treatment. Groups I to IV show AE/SAEs during the Core phase; Group V shows AE/SAEs during the Extension phase. During the Core phase, CV events being study endpoints were exempt from AE/SAE reporting; in contrast, during the Extension phase, all CV events were reported as AEs/SAEs.
Groups:
- Group V: Extension phase: Switched to open-label Canakinumab 150 mg quarterly subcutaneous + standard of care (SoC) therapy.
Arm/Group | Group I | Group II | Group III | Group IV | Group V
All-Cause Mortality (participants affected / at risk) | 239/2263 | 240/2285 | 228/2170 | 378/3348 | 211/5777
Serious Adverse Events (participants affected / at risk) | 759/2263 | 743/2285 | 686/2170 | 1099/3348 | 1216/5777
Other Adverse Events (participants affected / at risk) | 1271/2263 | 1324/2285 | 1199/2170 | 1905/3348 | 1497/5777
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group I (N=2263) | Group II (N=2285) | Group III (N=2170) | Group IV (N=3348) | Group V (N=5777)
Abnormal clotting factor (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 15 | 10 | 4 | 14 | 10
Bone marrow oedema (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 4 | 2 | 5 | 1 | 1
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Hilar lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 3 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 1
Monoclonal B-cell lymphocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 3 | 1
Polycythaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 1
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 0 | 3 | 3 | 0
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 6 | 1 | 4 | 4 | 14
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 2 | 2 | 2 | 7 | 71
Adams-Stokes syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 42 | 41 | 37 | 76 | 66
Angina unstable (Cardiac disorders) | 39 | 34 | 37 | 63 | 56
Aortic valve incompetence (Cardiac disorders) | 1 | 1 | 0 | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 3 | 2 | 2 | 3 | 2
Arrhythmia (Cardiac disorders) | 4 | 0 | 1 | 3 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 3 | 2
Arteriospasm coronary (Cardiac disorders) | 1 | 1 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 6 | 4 | 4 | 49
Atrial flutter (Cardiac disorders) | 2 | 0 | 1 | 1 | 6
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Atrial thrombosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Atrioventricular block (Cardiac disorders) | 0 | 1 | 1 | 2 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 1 | 2 | 4 | 4
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 4 | 2 | 4 | 2
Bradyarrhythmia (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 4 | 2 | 3 | 10 | 6
Cardiac aneurysm (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 2 | 7 | 7 | 15 | 9
Cardiac discomfort (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 5 | 4 | 7 | 4 | 43
Cardiac failure acute (Cardiac disorders) | 2 | 2 | 0 | 0 | 16
Cardiac failure chronic (Cardiac disorders) | 5 | 2 | 2 | 2 | 15
Cardiac failure congestive (Cardiac disorders) | 4 | 2 | 0 | 0 | 30
Cardiac fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac pseudoaneurysm (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 2 | 0 | 0 | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 2 | 2 | 3 | 1 | 6
Cardiogenic shock (Cardiac disorders) | 1 | 3 | 3 | 7 | 9
Cardiomegaly (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 1 | 1 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Conduction disorder (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cor pulmonale (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 9 | 10 | 5 | 20 | 27
Coronary artery insufficiency (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 1 | 0 | 1 | 3
Coronary artery stenosis (Cardiac disorders) | 2 | 1 | 0 | 2 | 14
Hypertensive heart disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Intracardiac thrombus (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 3 | 5 | 2 | 4 | 6
Left ventricular dysfunction (Cardiac disorders) | 2 | 0 | 0 | 1 | 3
Left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Microvascular coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 5 | 3 | 0 | 1 | 3
Myocardial infarction (Cardiac disorders) | 4 | 2 | 5 | 2 | 42
Myocardial ischaemia (Cardiac disorders) | 6 | 3 | 5 | 6 | 10
Nodal arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Palpitations (Cardiac disorders) | 3 | 2 | 2 | 1 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 2 | 1 | 0 | 2 | 0
Prinzmetal angina (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Pulseless electrical activity (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Right ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Right ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Silent myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
Sinus arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 3 | 0 | 2 | 2 | 1
Sinus node dysfunction (Cardiac disorders) | 4 | 2 | 5 | 4 | 6
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 3 | 1 | 1 | 2 | 1
Torsade de pointes (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
Trifascicular block (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 1 | 2 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 2 | 2 | 1
Ventricular fibrillation (Cardiac disorders) | 4 | 9 | 3 | 7 | 7
Ventricular tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 10 | 5 | 9 | 16 | 18
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0
Branchial cyst (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Cerebrovascular arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0
Hereditary haemochromatosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 1
Nonketotic hyperglycinaemia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0 | 0
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 2 | 0 | 0 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Otosclerosis (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Presbyacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 5 | 4 | 4 | 4
Vertigo positional (Ear and labyrinth disorders) | 2 | 2 | 3 | 2 | 2
Goitre (Endocrine disorders) | 1 | 0 | 1 | 2 | 0
Hyperparathyroidism primary (Endocrine disorders) | 1 | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 1 | 0
Hypopituitarism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 1 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Primary hyperaldosteronism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Toxic goitre (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Amaurosis fugax (Eye disorders) | 0 | 0 | 0 | 1 | 0
Angle closure glaucoma (Eye disorders) | 1 | 1 | 0 | 0 | 0
Blindness (Eye disorders) | 0 | 1 | 0 | 1 | 0
Blindness transient (Eye disorders) | 0 | 1 | 0 | 0 | 0
Blindness unilateral (Eye disorders) | 0 | 2 | 0 | 0 | 0
Cataract (Eye disorders) | 4 | 8 | 5 | 12 | 8
Cataract cortical (Eye disorders) | 1 | 0 | 0 | 0 | 0
Cataract diabetic (Eye disorders) | 0 | 1 | 0 | 0 | 0
Cataract nuclear (Eye disorders) | 0 | 1 | 0 | 0 | 0
Corneal degeneration (Eye disorders) | 1 | 0 | 0 | 0 | 0
Corneal infiltrates (Eye disorders) | 0 | 1 | 0 | 0 | 0
Dacryostenosis acquired (Eye disorders) | 2 | 0 | 0 | 0 | 0
Diabetic retinopathy (Eye disorders) | 0 | 0 | 0 | 2 | 1
Eye haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 1
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 2 | 0
Lens dislocation (Eye disorders) | 0 | 1 | 0 | 0 | 0
Macular degeneration (Eye disorders) | 0 | 0 | 1 | 0 | 0
Macular fibrosis (Eye disorders) | 0 | 0 | 0 | 1 | 0
Macular hole (Eye disorders) | 0 | 1 | 0 | 1 | 0
Macular oedema (Eye disorders) | 0 | 0 | 0 | 0 | 1
Neovascular age-related macular degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 1
Ocular ischaemic syndrome (Eye disorders) | 0 | 0 | 0 | 0 | 1
Papilloedema (Eye disorders) | 0 | 0 | 1 | 0 | 0
Retinal artery thrombosis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 2 | 2 | 0 | 2 | 2
Retinal haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0
Retinal vein occlusion (Eye disorders) | 0 | 0 | 0 | 0 | 1
Retinal vein thrombosis (Eye disorders) | 0 | 1 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 1 | 1 | 2
Abdominal adhesions (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 3 | 1 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 4 | 10 | 10 | 6
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 6 | 2 | 3 | 2 | 4
Acute abdomen (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Anal skin tags (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Anal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Anal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Anorectal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Appendiceal mucocoele (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Appendix disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 3 | 3 | 2 | 3 | 4
Colitis ischaemic (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 1
Colitis microscopic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 0
Colonic fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 2 | 1 | 4 | 3
Crohn's disease (Gastrointestinal disorders) | 1 | 3 | 1 | 2 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diabetic gastroenteropathy (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 5 | 4 | 2 | 3
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Duodenal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 2
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0
Duodenitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 2
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Erosive duodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Gallstone ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 0
Gastric ulcer (Gastrointestinal disorders) | 7 | 6 | 0 | 1 | 2
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Gastric volvulus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 4 | 1 | 4 | 6 | 4
Gastritis erosive (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastroduodenitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0
Gastrointestinal erosion (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 13 | 16 | 14 | 13 | 5
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal vascular malformation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 5 | 1 | 4 | 4
Haematemesis (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 3
Haematochezia (Gastrointestinal disorders) | 1 | 3 | 1 | 2 | 0
Haemorrhagic necrotic pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 3 | 1 | 2 | 1
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 2
Ileal ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Ileus (Gastrointestinal disorders) | 3 | 1 | 2 | 3 | 2
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2
Inguinal hernia (Gastrointestinal disorders) | 8 | 5 | 7 | 7 | 8
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Intestinal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Intestinal infarction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2
Intestinal mass (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1 | 3 | 2 | 2
Intestinal perforation (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 0
Intestinal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0
Ischaemic enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 3 | 4 | 2 | 12 | 6
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 4 | 1 | 0 | 2
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1
Melaena (Gastrointestinal disorders) | 2 | 1 | 0 | 2 | 3
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Mesenteric artery thrombosis (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0
Mesenteric vascular insufficiency (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Mouth cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Narcotic bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 3 | 2 | 4 | 0
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Oesophageal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oesophageal rupture (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatic disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pancreatic duct dilatation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pancreatic mass (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 6 | 6 | 3 | 11 | 3
Pancreatitis acute (Gastrointestinal disorders) | 3 | 6 | 2 | 3 | 6
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 2
Pancreatitis necrotising (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1
Peptic ulcer (Gastrointestinal disorders) | 2 | 0 | 0 | 3 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Ranula (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 6 | 1 | 1 | 3
Rectal lesion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Rectal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Rectal polyp (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Salivary gland calculus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 1 | 2 | 1 | 9
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Small intestine ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2
Subileus (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 4 | 2 | 4 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 8 | 8 | 8 | 3
Vomiting (Gastrointestinal disorders) | 5 | 4 | 2 | 4 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 4 | 2 | 1 | 3 | 3
Cardiac death (General disorders) | 0 | 0 | 0 | 0 | 4
Chest discomfort (General disorders) | 2 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 3 | 12 | 2 | 9 | 9
Chills (General disorders) | 1 | 1 | 0 | 0 | 0
Complication associated with device (General disorders) | 0 | 0 | 1 | 1 | 0
Death (General disorders) | 1 | 0 | 1 | 4 | 12
Drowning (General disorders) | 0 | 0 | 1 | 0 | 0
Drug intolerance (General disorders) | 0 | 0 | 0 | 0 | 1
Exercise tolerance decreased (General disorders) | 0 | 1 | 0 | 0 | 0
Facial pain (General disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 1 | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 2 | 2
Generalised oedema (General disorders) | 0 | 1 | 0 | 0 | 1
Hernia (General disorders) | 0 | 0 | 0 | 0 | 2
Heteroplasia (General disorders) | 0 | 0 | 0 | 0 | 1
Hyperplasia (General disorders) | 0 | 0 | 0 | 0 | 1
Hypothermia (General disorders) | 0 | 0 | 1 | 0 | 0
Impaired healing (General disorders) | 0 | 1 | 1 | 2 | 0
Implant site irritation (General disorders) | 0 | 1 | 0 | 0 | 0
Incarcerated hernia (General disorders) | 0 | 0 | 1 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 1 | 0
Ischaemic ulcer (General disorders) | 0 | 1 | 1 | 0 | 0
Local swelling (General disorders) | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 1 | 0 | 1 | 0
Mass (General disorders) | 0 | 1 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 3 | 2 | 0 | 3 | 6
Necrosis (General disorders) | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 44 | 48 | 39 | 75 | 35
Oedema peripheral (General disorders) | 2 | 0 | 1 | 3 | 1
Pacemaker syndrome (General disorders) | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0
Polyp (General disorders) | 0 | 0 | 1 | 0 | 0
Pseudocyst (General disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 4 | 4 | 6 | 5 | 3
Stent-graft endoleak (General disorders) | 0 | 0 | 1 | 1 | 1
Sudden cardiac death (General disorders) | 0 | 1 | 1 | 0 | 11
Sudden death (General disorders) | 0 | 0 | 0 | 1 | 7
Surgical failure (General disorders) | 0 | 0 | 1 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 3 | 2 | 0
Vascular stent restenosis (General disorders) | 2 | 2 | 1 | 1 | 0
Vascular stent stenosis (General disorders) | 0 | 0 | 1 | 0 | 3
Vascular stent thrombosis (General disorders) | 0 | 1 | 0 | 0 | 0
Vessel puncture site haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 0
Alcoholic liver disease (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 2 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 4 | 0 | 1 | 2 | 1
Biliary cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1
Biliary fistula (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 2 | 4 | 0 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 1 | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 11 | 4 | 8 | 9 | 7
Cholecystitis acute (Hepatobiliary disorders) | 5 | 7 | 4 | 7 | 5
Cholelithiasis (Hepatobiliary disorders) | 8 | 8 | 8 | 18 | 4
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 1 | 0 | 0
Gallbladder polyp (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Haemorrhagic hepatic cyst (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 4
Hepatic congestion (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Hepatic vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hepatorenal failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hydrocholecystis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 2
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Non-alcoholic fatty liver (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Steatohepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Allergy to arthropod sting (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 1 | 0 | 0 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0 | 1 | 2
Contrast media allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 2 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 2 | 0 | 0 | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Abdominal sepsis (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Abscess intestinal (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Abscess jaw (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Abscess limb (Infections and infestations) | 4 | 1 | 3 | 3 | 0
Abscess neck (Infections and infestations) | 1 | 0 | 0 | 2 | 0
Abscess oral (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Abscess soft tissue (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Acute hepatitis B (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 1 | 1 | 2 | 2
Appendicitis (Infections and infestations) | 3 | 4 | 6 | 4 | 3
Appendicitis perforated (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 1 | 0 | 1 | 1
Arthritis infective (Infections and infestations) | 1 | 0 | 0 | 3 | 1
Atypical pneumonia (Infections and infestations) | 0 | 2 | 0 | 2 | 0
Bacteraemia (Infections and infestations) | 3 | 1 | 1 | 1 | 2
Bacterial disease carrier (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Bacterial sepsis (Infections and infestations) | 1 | 2 | 0 | 0 | 0
Bacteroides infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bartholin's abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bone abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 10 | 9 | 6 | 14 | 10
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 1 | 2 | 0
Bursitis infective (Infections and infestations) | 0 | 1 | 1 | 1 | 1
Bursitis infective staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Campylobacter gastroenteritis (Infections and infestations) | 2 | 0 | 1 | 0 | 0
Campylobacter infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Carbuncle (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 29 | 32 | 19 | 27 | 22
Cellulitis gangrenous (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cellulitis of male external genital organ (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cellulitis staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Central nervous system infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Chikungunya virus infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Cholangitis infective (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0 | 0 | 1 | 1
Chorioretinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Chronic tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Clostridial infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 3 | 1 | 4 | 1 | 1
Clostridium difficile infection (Infections and infestations) | 2 | 1 | 2 | 1 | 0
Colonic abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Creutzfeldt-Jakob disease (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 2 | 0 | 3 | 1 | 1
Dengue fever (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 2 | 4 | 1
Device related sepsis (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Diabetic foot infection (Infections and infestations) | 2 | 0 | 0 | 1 | 2
Diabetic gangrene (Infections and infestations) | 0 | 0 | 1 | 2 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 8 | 9 | 8 | 13 | 6
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Empyema (Infections and infestations) | 2 | 0 | 1 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 1 | 2 | 2 | 1
Endocarditis bacterial (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 3 | 2 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Epiglottitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 6 | 12 | 6 | 9 | 13
Escherichia sepsis (Infections and infestations) | 0 | 1 | 2 | 3 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1
External ear cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gallbladder abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gallbladder empyema (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gangrene (Infections and infestations) | 1 | 1 | 5 | 0 | 2
Gastritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 6 | 5 | 6 | 8 | 4
Gastroenteritis clostridial (Infections and infestations) | 2 | 0 | 1 | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 2 | 0 | 2 | 1 | 0
Gastrointestinal bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Groin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Haematoma infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Haemophilus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Haemophilus sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Haemorrhagic pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Helicobacter infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Hepatic amoebiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Hepatitis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes ophthalmic (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 4 | 1
Human ehrlichiosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hypopyon (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Implant site abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Implant site infection (Infections and infestations) | 0 | 1 | 2 | 0 | 1
Incision site cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Incision site infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infected bite (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Infected cyst (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Infectious colitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 3 | 1 | 0 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 5 | 0 | 2 | 3 | 1
Infective spondylitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 4 | 6 | 2 | 3 | 9
Intervertebral discitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Joint abscess (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Labyrinthitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Leptospirosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Localised infection (Infections and infestations) | 2 | 2 | 3 | 5 | 4
Lower respiratory tract infection (Infections and infestations) | 3 | 2 | 4 | 4 | 4
Lung abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 2 | 0 | 3 | 1 | 1
Lyme disease (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Malaria (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Mastoiditis (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Mediastinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Medical device site infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Meningitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Meningitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Meningococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Mesenteric abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Metapneumovirus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Muscle abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Mycobacterial infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Mycobacterium avium complex infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 2 | 1 | 1 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Orchitis (Infections and infestations) | 1 | 0 | 2 | 0 | 0
Osteomyelitis (Infections and infestations) | 4 | 3 | 3 | 4 | 10
Osteomyelitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Osteomyelitis blastomyces (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1 | 2 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Otitis media acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Otitis media chronic (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pancreatic abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Parametritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Parotitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Pelvic abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Perichondritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Perineal abscess (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Periodontitis (Infections and infestations) | 1 | 1 | 0 | 2 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 2 | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Peritoneal abscess (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 2 | 1 | 3 | 2 | 2
Pharyngeal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pilonidal cyst (Infections and infestations) | 1 | 0 | 0 | 0 | 2
Pneumococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 67 | 60 | 53 | 83 | 70
Pneumonia bacterial (Infections and infestations) | 1 | 1 | 0 | 3 | 1
Pneumonia escherichia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia haemophilus (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia legionella (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Pneumonia necrotising (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Pneumonia pseudomonal (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Post procedural cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Post procedural infection (Infections and infestations) | 1 | 2 | 0 | 0 | 4
Post procedural sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Postoperative abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Postoperative wound infection (Infections and infestations) | 2 | 2 | 2 | 1 | 4
Proctitis infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Propionibacterium infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pseudomembranous colitis (Infections and infestations) | 1 | 0 | 2 | 0 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pseudomonas bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Psoas abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 2 | 2 | 1 | 2
Pulmonary tuberculosis (Infections and infestations) | 1 | 2 | 1 | 1 | 0
Pyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 3 | 1 | 2 | 5 | 2
Pyelonephritis acute (Infections and infestations) | 1 | 5 | 1 | 3 | 0
Pyoderma (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pyuria (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Renal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 3
Respiratory tract infection (Infections and infestations) | 2 | 7 | 0 | 7 | 2
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Rubella (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Salmonellosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Scrotal abscess (Infections and infestations) | 1 | 0 | 1 | 1 | 0
Scrub typhus (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Sepsis (Infections and infestations) | 19 | 25 | 15 | 19 | 22
Sepsis syndrome (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Septic embolus (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Septic necrosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 6 | 8 | 6 | 11 | 3
Sialoadenitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 3 | 1 | 0 | 2 | 3
Sinusitis fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Staphylococcal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 2 | 1 | 0 | 0 | 3
Staphylococcal infection (Infections and infestations) | 1 | 1 | 2 | 1 | 2
Staphylococcal mediastinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 1 | 2 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 2 | 0
Streptococcal sepsis (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 4 | 3 | 2 | 3 | 0
Subdiaphragmatic abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Subdural empyema (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Testicular abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tetanus (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 1 | 1 | 1
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 13 | 11 | 10 | 21 | 19
Urinary tract infection bacterial (Infections and infestations) | 3 | 0 | 1 | 0 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection fungal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 4 | 4 | 5 | 3 | 7
Vestibular neuronitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Viral cardiomyopathy (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Viral diarrhoea (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Vulval abscess (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 3 | 4 | 0 | 2
Wound infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Wound sepsis (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 5 | 0 | 3 | 4 | 4
Arterial injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Asbestosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Central cord syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 2 | 2
Chest injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2 | 2
Closed globe injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 3 | 5 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0
Dural tear (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 1 | 2 | 3 | 9
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 5 | 2 | 5 | 2
Femur fracture (Injury, poisoning and procedural complications) | 1 | 3 | 2 | 5 | 4
Foot fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 1 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Gallbladder injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Gastrointestinal stoma necrosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 3 | 2
Hip fracture (Injury, poisoning and procedural complications) | 1 | 2 | 3 | 6 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 4 | 2
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 3 | 2
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Intentional product misuse (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 4 | 0 | 3 | 3 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 0 | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 3 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 3 | 2
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 3 | 5 | 8 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Muscle contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 0
Musculoskeletal foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 1 | 2 | 2 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 1 | 0
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Pneumoconiosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Post procedural fever (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 3 | 0
Postoperative hernia (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0
Procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Radiation mucositis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 3 | 1
Rib fracture (Injury, poisoning and procedural complications) | 4 | 3 | 3 | 7 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 4 | 1 | 2 | 3 | 3
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 5 | 1
Spinal cord injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
Stab wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 2 | 2 | 1 | 2 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 4 | 4 | 5 | 5
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 4 | 2 | 0 | 0 | 2
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 3 | 2
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 2 | 0
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Traumatic amputation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Traumatic arthritis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 3 | 2
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Vascular graft complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Anticoagulation drug level above therapeutic (Investigations) | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood creatine phosphokinase MB increased (Investigations) | 0 | 1 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood urine present (Investigations) | 0 | 1 | 0 | 0 | 0
Body mass index decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Central venous pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0
Chest X-ray abnormal (Investigations) | 0 | 0 | 0 | 2 | 0
Clostridium test positive (Investigations) | 0 | 0 | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 1 | 1 | 1 | 1 | 0
Haemoglobin decreased (Investigations) | 2 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 3 | 0
Human metapneumovirus test positive (Investigations) | 0 | 0 | 0 | 0 | 1
Imaging procedure abnormal (Investigations) | 0 | 0 | 1 | 0 | 0
International normalised ratio decreased (Investigations) | 0 | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 0 | 1 | 1 | 0
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Quality of life decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Scan myocardial perfusion abnormal (Investigations) | 0 | 0 | 0 | 0 | 2
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 1
Troponin increased (Investigations) | 1 | 1 | 0 | 1 | 2
Volume blood decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 2
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 6 | 6 | 6 | 8
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 10 | 1 | 11 | 8
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 1 | 7 | 3 | 1
Diabetes with hyperosmolarity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Diabetic complication (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 2 | 1 | 1 | 0
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 4 | 3 | 6 | 4
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 4 | 3 | 3 | 7
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 4 | 3 | 9 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 9 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 4 | 2 | 4
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1 | 0
Insulin resistant diabetes (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Insulin-requiring type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 2 | 2 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 5 | 1 | 1 | 2 | 4
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 | 2 | 1 | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 2 | 4 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 3 | 2
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 8 | 5 | 7 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 4 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3
Chondromalacia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Finger deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0
Fracture malunion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Gouty tophus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 0
Immunoglobulin G4 related disease (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Intervertebral disc calcification (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 3 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 2 | 6 | 10 | 6
Jaw cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1 | 5 | 5
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0
Muscle swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 5 | 5 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 4 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 0
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 2
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 19 | 21 | 18 | 51 | 26
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 1 | 1 | 2 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 3 | 3
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 5 | 3
Shoulder deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 6 | 2 | 4 | 4 | 4
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3 | 5 | 3
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Vertebral wedging (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 3 | 2 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 2 | 3 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 2 | 5 | 3
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Adenosquamous cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 1
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1 | 0
Angiolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 2 | 0
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 | 18 | 18 | 21 | 30
Benign cardiac neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Benign neoplasm of scrotum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Benign small intestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Benign urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5 | 3 | 5 | 2
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 3
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 2 | 0 | 0
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 2 | 3 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 5 | 2 | 4
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Brenner tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 3 | 3
Carcinoid tumour of the gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 0 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1 | 2
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4 | 5 | 6 | 3
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Diffuse large B-cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Ductal adenocarcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Endometrial cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1 | 1 | 5 | 5
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 3 | 0
Hepatic cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1 | 2 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0
Inflammatory pseudotumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 2 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 3 | 0
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 3 | 7 | 1
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 1 | 0
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Lung carcinoma cell type unspecified stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 9 | 9 | 25 | 14
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 1 | 0
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Malignant fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Malignant mediastinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5 | 3 | 2 | 4
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 2 | 0 | 1
Malignant neoplasm of pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 2
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 2 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 1 | 1
Metastases to kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5 | 1 | 4 | 2
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 5 | 2 | 2
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 1 | 0
Metastases to pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Metastases to rectum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1 | 0 | 0
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Mucinous adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Nasal cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 3 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0
Neuroendocrine breast tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 3 | 0
Non-Hodgkin's lymphoma refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 3 | 1 | 3
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Non-small cell lung cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 2 | 1
Oesophageal adenocarcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 4 | 2 | 2
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Oligodendroglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 3 | 5 | 3
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 3 | 0
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 2 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 2 | 2
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 1
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Pharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 2 | 0
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 10 | 10 | 13 | 15
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 0 | 1
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2 | 2 | 3 | 1
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 3 | 2 | 1
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 5 | 1 | 3
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0
Rosai-Dorfman syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 5 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Small intestine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 5 | 6 | 10 | 9
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5 | 0 | 2 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 1 | 3 | 1
Squamous cell carcinoma of the hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Superficial spreading melanoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Thyroid cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0
Tonsil cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 4
Transitional cell carcinoma urethra (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 2
Amnesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Apraxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Brain injury (Nervous system disorders) | 0 | 3 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Carotid artery aneurysm (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Carotid artery disease (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 1 | 1 | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 3 | 0 | 2 | 1 | 8
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 1 | 0 | 3
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cerebellar infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cerebellar stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Cerebral arteriosclerosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 2
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 9
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1 | 0 | 3
Cerebrovascular accident (Nervous system disorders) | 2 | 1 | 1 | 4 | 22
Cervical myelopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Coma (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Dementia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Dementia Alzheimer's type (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dementia with Lewy bodies (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Diabetic coma (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Diplegia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 6 | 2 | 3 | 7 | 4
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 2 | 0 | 0 | 0 | 1
Dystonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 1 | 3
Epilepsy (Nervous system disorders) | 2 | 2 | 1 | 1 | 2
Facial paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Focal dyscognitive seizures (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 1 | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhagic transformation stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 4 | 3 | 3 | 4 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypersomnia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 2 | 1
Hypoglycaemic coma (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 2
IIIrd nerve paresis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 16
Lacunar infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Lacunar stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 3 | 0 | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 2
Lumbosacral radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Mental impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 1 | 0 | 2 | 1
Migraine (Nervous system disorders) | 1 | 1 | 0 | 1 | 2
Mixed dementia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Orthostatic intolerance (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Paresis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Peripheral nerve lesion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0 | 1 | 1
Post herpetic neuralgia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Post stroke seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 2 | 1 | 2 | 4 | 2
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 5 | 4 | 0
Seizure (Nervous system disorders) | 3 | 2 | 1 | 4 | 2
Sensory disturbance (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Spinal claudication (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Spinal cord infarction (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Spondylitic myelopathy (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Stupor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Subdural hygroma (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 15 | 17 | 16 | 25 | 16
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Thalamic infarction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Thrombotic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Tonic convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Transient global amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1 | 0 | 15
Trigeminal neuralgia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0
Upper motor neurone lesion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
VIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Vascular dementia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Vascular encephalopathy (Nervous system disorders) | 0 | 2 | 0 | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0 | 1 | 0 | 1
Device battery issue (Product Issues) | 2 | 0 | 2 | 0 | 1
Device dislocation (Product Issues) | 0 | 1 | 2 | 1 | 1
Device end of service (Product Issues) | 0 | 1 | 1 | 0 | 0
Device failure (Product Issues) | 1 | 0 | 1 | 0 | 0
Device inappropriate shock delivery (Product Issues) | 0 | 0 | 1 | 0 | 0
Device issue (Product Issues) | 0 | 0 | 1 | 0 | 0
Device lead damage (Product Issues) | 0 | 0 | 0 | 1 | 0
Device lead issue (Product Issues) | 0 | 0 | 0 | 1 | 0
Device loosening (Product Issues) | 1 | 0 | 0 | 1 | 0
Device malfunction (Product Issues) | 1 | 2 | 1 | 3 | 0
Device occlusion (Product Issues) | 0 | 0 | 0 | 1 | 0
Device signal detection issue (Product Issues) | 0 | 0 | 0 | 0 | 1
Lead dislodgement (Product Issues) | 0 | 0 | 1 | 0 | 0
Acute stress disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Adjustment disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Affective disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Alcoholic psychosis (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Alcoholism (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 3 | 2
Anxiety disorder (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0
Anxiety disorder due to a general medical condition (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Bipolar I disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0
Burnout syndrome (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1 | 1
Conversion disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 2 | 1 | 2 | 2
Delirium tremens (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 7 | 4 | 2 | 4 | 2
Dissociative amnesia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Drug use disorder (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Generalised anxiety disorder (Psychiatric disorders) | 2 | 1 | 0 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Head banging (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Homicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Major depression (Psychiatric disorders) | 2 | 1 | 1 | 1 | 0
Mental status changes (Psychiatric disorders) | 4 | 0 | 2 | 6 | 2
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Schizophrenia (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0
Somnambulism (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 1 | 1 | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 20 | 30 | 16 | 27 | 22
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Anuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Calculus bladder (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 3
Calculus urethral (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 4 | 5 | 4 | 4 | 5
Diabetic nephropathy (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1
End stage renal disease (Renal and urinary disorders) | 1 | 1 | 0 | 2 | 1
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Glomerulonephritis membranous (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 5 | 6 | 3 | 7 | 3
Hydronephrosis (Renal and urinary disorders) | 2 | 3 | 1 | 2 | 0
Hypertensive nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Lower urinary tract symptoms (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 3 | 2 | 4 | 7 | 3
Nephrotic syndrome (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Prerenal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Renal artery stenosis (Renal and urinary disorders) | 1 | 0 | 0 | 2 | 1
Renal artery thrombosis (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 2 | 0 | 2 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 7 | 10 | 11 | 13 | 5
Renal haematoma (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 4 | 3 | 1 | 4
Renal injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
Renal mass (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 1 | 2 | 7 | 3
Urethral obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urinary bladder polyp (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 4 | 4 | 3 | 4 | 6
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 1
Vesicocutaneous fistula (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 5 | 6 | 5 | 5 | 8
Cystocele (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Epididymal cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Genital atrophy (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Genital prolapse (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 2 | 1 | 0 | 1 | 0
Prostatic haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Prostatic mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Prostatism (Reproductive system and breast disorders) | 0 | 1 | 1 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 2 | 0 | 2 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 2 | 1 | 1 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Spermatocele (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0
Uterine cervix stenosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Varicocele (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Varicose veins pelvic (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 4 | 4 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 | 7 | 11 | 13 | 21
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 0 | 3 | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 3 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 1
Cheyne-Stokes respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 28 | 21 | 16 | 40 | 33
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 | 8 | 10 | 23 | 19
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 1 | 1
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2 | 6 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 4 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 3 | 5
Idiopathic interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 2 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Lung hernia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pleural adhesion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 4 | 6 | 4
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0 | 3 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0 | 4 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 2 | 18
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 4 | 1
Pulmonary haematoma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 3
Pulmonary microemboli (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 1 | 2 | 5
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 12 | 11 | 9 | 12 | 5
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 5 | 2
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Vocal cord leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 3 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Brow ptosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 6 | 1 | 0 | 4
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 1
Rhinophyma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 5 | 5 | 3 | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Homicide (Social circumstances) | 0 | 1 | 0 | 0 | 0
Accelerated hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Aneurysm ruptured (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Angiodysplasia (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 8 | 4 | 6 | 6 | 12
Aortic aneurysm rupture (Vascular disorders) | 0 | 1 | 0 | 0 | 3
Aortic dissection (Vascular disorders) | 0 | 0 | 1 | 0 | 2
Aortic stenosis (Vascular disorders) | 1 | 0 | 2 | 0 | 1
Aortitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Arterial haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Arterial insufficiency (Vascular disorders) | 0 | 0 | 1 | 1 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0 | 2 | 5
Arteriovenous fistula (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Arteritis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Brachiocephalic artery stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Circulatory collapse (Vascular disorders) | 3 | 1 | 3 | 1 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 5
Embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Embolism arterial (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Embolism venous (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Essential hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1 | 1 | 2 | 2
Femoral artery aneurysm (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Femoral artery embolism (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 2 | 3 | 1 | 5 | 5
Haemodynamic instability (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 10 | 8 | 8 | 15 | 17
Hypertensive crisis (Vascular disorders) | 7 | 5 | 2 | 11 | 5
Hypertensive emergency (Vascular disorders) | 1 | 2 | 1 | 0 | 1
Hypotension (Vascular disorders) | 8 | 5 | 4 | 11 | 6
Hypovolaemic shock (Vascular disorders) | 2 | 1 | 0 | 0 | 1
Intermittent claudication (Vascular disorders) | 1 | 1 | 0 | 3 | 3
Internal haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Ischaemic limb pain (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Lymphatic fistula (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Lymphorrhoea (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Malignant hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Orthostatic hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 3 | 1 | 0 | 2
Pallor (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 3 | 4 | 2 | 4 | 11
Peripheral artery aneurysm (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 3 | 2 | 0 | 4
Peripheral artery stenosis (Vascular disorders) | 1 | 2 | 1 | 1 | 6
Peripheral artery thrombosis (Vascular disorders) | 0 | 2 | 1 | 1 | 1
Peripheral embolism (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 11
Peripheral vascular disorder (Vascular disorders) | 0 | 3 | 2 | 1 | 4
Peripheral venous disease (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Shock (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Temporal arteritis (Vascular disorders) | 1 | 0 | 1 | 1 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Varicose ulceration (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 1 | 0 | 0
Vascular insufficiency (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group I (N=2263) | Group II (N=2285) | Group III (N=2170) | Group IV (N=3348) | Group V (N=5777)
Angina pectoris (Cardiac disorders) | 142 | 164 | 129 | 228 | 115
Diarrhoea (Gastrointestinal disorders) | 138 | 146 | 137 | 216 | 110
Fatigue (General disorders) | 113 | 99 | 84 | 169 | 72
Non-cardiac chest pain (General disorders) | 142 | 143 | 111 | 228 | 68
Oedema peripheral (General disorders) | 136 | 142 | 134 | 173 | 110
Bronchitis (Infections and infestations) | 131 | 162 | 114 | 234 | 160
Influenza (Infections and infestations) | 141 | 145 | 118 | 194 | 154
Upper respiratory tract infection (Infections and infestations) | 153 | 156 | 134 | 252 | 125
Urinary tract infection (Infections and infestations) | 126 | 129 | 93 | 175 | 123
Viral upper respiratory tract infection (Infections and infestations) | 264 | 297 | 263 | 388 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 165 | 181 | 144 | 252 | 184
Back pain (Musculoskeletal and connective tissue disorders) | 169 | 177 | 157 | 277 | 163
Pain in extremity (Musculoskeletal and connective tissue disorders) | 145 | 145 | 98 | 204 | 128
Dizziness (Nervous system disorders) | 114 | 126 | 132 | 189 | 107
Headache (Nervous system disorders) | 133 | 111 | 120 | 178 | 72
Cough (Respiratory, thoracic and mediastinal disorders) | 151 | 152 | 121 | 233 | 103
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 126 | 123 | 110 | 193 | 112
Hypertension (Vascular disorders) | 198 | 216 | 208 | 309 | 241

LIMITATIONS AND CAVEATS:
Comparison across groups is no longer feasible in the Extension phase because all patients received canakinumab 150 mg. Beyond the primary endpoint, all p-values for the canakinumab 50 mg and 300 mg groups are to be considered nominal only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-09-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT01327846/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-14): https://cdn.clinicaltrials.gov/large-docs/46/NCT01327846/SAP_001.pdf